| MD Anderson IND Sponsor Cover Sheet | |
|---|---|
| Protocol ID | 2016-0250 |
| Protocol Title | Phase 1 Study of IACS-010759 in Subjects with Relapsed or Refractory AML |
| Protocol Phase | 1 |
| Protocol Version | 11 |
| Version Date | January 21, 2020 |
| Protocol PI | Marina Konopleva, M.D. |
| Department | Leukemia |
| IND Sponsor | MD Anderson Cancer Center |
| IND# | 128,639 |

| Study Protocol: IACS2015-001 | MDACC Protocol ID: 2016-0250 |
|------------------------------|------------------------------|
| Version: Amendment #11 | Version Date: 01-21-20 |

## Phase 1 Study of IACS-010759 in Subjects with relapsed or refractory AML

#### Study Synopsis and Objectives

This is an open label Phase 1 study of IACS-10579 utilizing a 3+3 dose-escalation phase followed by an expansion phase in subjects with relapsed or refractory AML and no available treatment options with known benefit.

In cohorts 1 and 2, in the first cycle, IACS-010759 will be administered on Day 1 followed by continuous dosing starting on day 8 through day 28; cycles 2 and beyond will be continuous daily dosing. Based on PK analysis and modeling of preliminary data from cohorts 1 and 2, the study design has been amended. In cohort 3 and subsequent cohorts, in the first cycle, IACS-010759 will be administered daily for up to 7 days during an initial Induction Phase (Day 1-7) followed the Maintenance Phase (Day 8-21), which will use a lower dose to maintain steady state drug levels. For cohort 3, the maintenance dose will be administered once weekly on Day 8 and Day 15 of the 21-day cycle in cycle 1; in subsequent cycles, doses will be administered on Days 1, 8 and 15 of each cycle, unless alternate schedules are recommended by the SMC. In subsequent cohorts, the induction and maintenance doses and/or the dosing interval during the maintenance phase may be further modified by the SMC based on safety, PK and PD data observed. Dosing will continue until confirmed progressive disease, initiation of alternative cancer therapy, unacceptable toxicity, or other reasons to discontinue treatment prematurely at the dose levels given below:

Original Dose Escalation Regimen, Cohorts 1 and 2:

| PHASE | COHORT | NO OF SUBJECTS | IACS-010759 DOSE LEVEL<br>(DAILY EXCEPT<br>CYCLE 1, DAY 2-7)<br>* |
|---|---|---|---|
| Dose- | Cohort 1 | 3-6 | 0.5 mg |
| escalation | Cohort 2 | 3-6 | 1 mg |

<sup>\*</sup>Intermediate doses of IACS-010759, not to exceed 8 mg, not listed above may also be pursued with SMC approval depending on the safety, PK and PD data observed.

#### Revised Dose Escalation Regimen for Cohorts 3-6 and Expansion Regimen for Cohort 7:

| DUACE | COLLORT | NO OF | INDUCTION DOSE* | MAINTENANCE DOSE* |
|---|---|---|---|---|
| PHASE | COHORT | SUBJECTS | (FREQUENCY#) | (FREQUENCY) |
| | Cohort 3 | 3-6 | 2 mg (daily, Cycle 1 Day 1-7) | 0.5 mg (once per week) |
| Dose- | Cohort 4** | 3-6 | 2.5 mg (daily, Cycle 1 Day 1-7) | 1.0 mg (three times per week) |
| escalation | Cohort 5 | 3-6 | 2.5 mg (daily, Cycle 1 Day 1-5) | 1.5 mg (three times per week) |
| | Cohort 6 | 3-6 | 3 mg (daily, Cycle 1 Day 1-5) | 2 mg (three times per week) |
| Expansion | Cohort 7 | 12 | RP2D | RP2D |

<sup>\*</sup>Intermediate induction or maintenance doses of IACS-010759, not to exceed 6 mg, and #alternative duration of induction doses or other maintenance schedules not listed above may also be pursued with SMC approval depending on the safety, PK and PD data observed.


Induction dose: 2.5 mg, administered daily, Cycle 1 Day 1 through Day 7

<sup>\*\*</sup>Following their review of Cohort 3, the SMC recommended implementation of the following dose schedule for subjects who enroll in Cohort 4 of the study:

## Phase 1 Study of IACS-010759 in Subjects with relapsed or refractory AML

#### **Study Synopsis and Objectives**

Maintenance dose: 1 mg, administered 3x/week (for a total weekly dose of 3 mg) with the first maintenance dose starting on Cycle 1 Day 8

Subjects in the expansion phase will be treated at the recommended phase 2 dose (RP2D) identified in the dose-escalation phase, using the induction + maintenance regimen.

Up to 48 subjects will be enrolled in the study: a maximum of 36 subjects in the dose-escalation and a maximum of 18 subjects in the expansion phase (12 additional subjects and the 6 subjects from the dose-escalation phase at the cohort of the highest dose level shown to be well tolerated or the recommended phase 2 dose).

The primary objective is to determine safety and tolerability of IACS-010759, the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D).

The secondary objectives are IACS-010759 pharmacokinetics, food effect, and preliminary clinical efficacy (overall response rates, duration of response, progression-free survival, overall survival).

The exploratory objective is to evaluate pharmacodynamic (PD) and exploratory biomarkers of activity of IACS-010759.

## **Table of Contents**

| 1 | Protocol | Amendments | 6 |
|---|---|---|---|
| 2 | Backgrou | und Information | 14 |
| | 2.1 AML | | 14 |
| | 2.2 IACS | i-010579 | 14 |
| | 2.2.1 | IACS-010759 Preclinical Biology | |
| | 2.2.2 | IACS-010759 Nonclinical Experience | |
| | 2.2.3 | IACS-010759 Chemical Properties | |
| 3 | Study Ra | tionale | 17 |
| | 3.1 Ratio | onale for IACS-010759 Dose Selection | 17 |
| | 3.2 Ratio | onale for Study Design | 18 |
| 4 | | ental Plan | |
| | • | ly Design | |
| | 4.1.1 | Study Phase | |
| | 4.1.2 | Enrollment/Randomization | |
| | 4.1.3 | Subject Population | |
| | 4.1.4 | Number of Sites and Subjects | |
| | 4.1.5 | Sample Size Considerations | |
| | 4.1.6 | Treatment Cohorts and Treatment Schema | |
| | 4.1.7 | Dose-escalation | 20 |
| | 4.1.8 | Expansion Phase | 21 |
| | 4.1.9 | Dosing Adjustments, Delays and Discontinuations | |
| | 4.1.9. | I IACS-010759 Dose Adjustments for Drug-Related Hematological AEs | 22 |
| | 4.1.9.2 | 2 IACS-010759 Dose adjustments for Non-Hematologic Drug-Related AEs | 23 |
| | 4.1.9.3 | | |
| | 4.1.9. | | |
| | 4.1.10 | DLT, MTD and RP2D definitions | |
| | 4.1.11 | Assessment of Elevated Lactic Acid Levels | |
| | 4.1.12 | Subject Withdrawal | |
| | 4.1.13 | Subject Evaluability and Replacement | |
| | 4.1.14 | Safety Monitoring and Study Stopping Rules | |
| | | .1 Study Stopping Rules | |
| | | .2 Protocol Violations and Deviations | |
| | 4.1.15 | Follow-Up at Treatment Discontinuation or Early Withdrawal | |
| | 4.1.16 | Long-Term Follow-Up | |
| | | ly Flowcharts | |
| | | ty and tolerability | |
| | 4.3.1 | Endpoints & Assessment Methods | |
| | 4.3.2 | Subject Evaluation & Statistics | |
| | | cal Efficacy | |
| | 4.4.1 | Subject Evaluation & Statistics | . 39 |

| | 4.4. | 2 | Endpoints & Assessment Methods | . 39 |
|---|---|---|---|---|
| | 4.5 | IACS | -010759 Plasma Drug Levels | . 40 |
| | 4.5. | 1 | Subject Evaluation & Statistics | . 40 |
| | 4.5. | 2 | Endpoints & Assessment Methods | . 41 |
| | 4.6 | Biolo | ogical activity of IACS-010759 | . 41 |
| | 4.6. | 1 | Subject Evaluation & Statistics | . 41 |
| | 4.6. | 2 | Endpoints & Assessment Methods | . 41 |
| 5 | Sub | ject E | ligibility | . 41 |
| | 5.1 | Inclu | sion Criteria | . 41 |
| | 5.2 | Exclu | usion Criteria | . 44 |
| 6 | Stud | dy Dr | ug | . 45 |
| | 6.1 | Stud | y Drug Administration | . 45 |
| | 6.2 | Stud | y Drug Information | . 46 |
| | 6.3 | Drug | Overdose Management | . 46 |
| 7 | Con | curre | nt and Supportive Therapies | . 47 |
| | 7.1 | Non | -Permitted Concomitant Therapies | . 47 |
| | 7.2 | Supp | portive Care Guidelines & Permitted Concomitant Therapies | . 47 |
| | 7.2. | | Concomitant medication/therapies | |
| | 7.2. | 2 | Use of Blood Products | . 48 |
| | 7.2. | 3 | Lactic Acidosis and Severe Acidemia Management | . 49 |
| 8 | Adn | ninist | rative, Legal & Ethical Requirements | . 49 |
| | 8.1 | Adve | erse Event, serious adverse event and reporting | . 49 |
| | 8.1. | 1 | Adverse Event (AE): | . 49 |
| | 8.1. | 2 | Reporting of Adverse Events | . 50 |
| | 8.1. | 3 | Assessing Severity of Adverse Events | . 50 |
| | 8.1. | 4 | Assessing Relationship to Study Treatment | |
| | 8.1. | 5 | Classification of Causality | |
| | 8.1. | | Reporting Requirements | |
| | 8.1. | - | Serious Adverse Event Reporting (SAE) | |
| | 8.1. | _ | Reporting to FDA: | |
| ^ | 8.1. | | Unexpected Adverse Event | |
| 9 | | | ces | |
| | 9.1 | | ses of elevated lactate | |
| | 9.2 | | of abbreviations | |
| | 9.3 | | G Performance Status* | |
| | 9.4 | | York Heart Association (NYHA) Functional Classification | |
| | 9.5 | Refe | rences | . 57 |

## 1 Protocol Amendments

| Section | Text | Amendments | Rationale for Change |
|---|---|---|---|
| | | Amendment #10<br>(dated 21 January 2019) | |
| Synopsis, 3.1,<br>4.1.6, 4.1.7, 4.2 | Revised | Revised the induction phase duration from 7 days to up to 7 days | SMC recommendation at<br>end of cohort 4 to reduce<br>the daily induction phase<br>dosing from 7 days to 5<br>days starting in cohort 5 |
| Synopsis, 4.1.6 | Revised | Modified the cohort 5 dosing regimen to 2.5 mg induction (daily, Cycle 1 Day 1 through Day 5) and 1.5 mg maintenance (3 times per week starting on Cycle 1 Day 8) | SMC recommendation |
| Synopsis, 4.1.6 | Revised | Modified the cohort 6 dosing regimen to 3 mg induction (daily, Cycle 1 Day 1 through Day 5) and 2 mg maintenance (3 times per week starting on Cycle 1 Day 8) | Original dose regimen for cohort 6 not likely to be tolerated based on available interim data |
| 4.2 | Revised | Changed Cycle 1 Day 7 visit to Cycle 1 Day 5 visit starting with subjects enrolled in cohort 5 | Collection of PK data<br>based on revised dosing<br>regimen |
| 4.2 | Added | Added PK assessment 24 hours post study drug administration on Cycle 1 Day 5 starting with subjects enrolled in cohort 5 | Revised dosing regimen |
| 4.2 | Removed | Removed days allowable for Cycle 1 Day 5 and Cycle 1 Day 8 | Consistency of PK data based on revised dosing regimen |
| Throughout | Clarification | Corrected typographical errors | Consistency and readability of protocol |
| | • | Amendment #9<br>(dated 13 September 2018) | |
| 4.2 | Added | Added baseline dilated eye exam with fundus photos and neurology & exam (prior to Cycle 1 Day 1 study drug administration) | SMC recommendation |
| 5.2 | Added | Updated eligibility to exclude patients with ≥ grade 1 peripheral neuropathy | SMC recommendation |
| | | Amendment #8<br>(dated 06 June 2018) | |
| 4.1.3, 5.1 | Removed | Removed eligibility requirement that subjects must have failed to achieve CR to standard induction therapy | Increased flexibility at site<br>based on available subject<br>safety information from<br>this study and ongoing<br>solid tumor study<br>(IACS2016-002) |
| | • | Amendment #7 | |
| | | (dated 27 February 2018) | |

| Section | Text | Amendments | Rationale for Change |
|---|---|---|---|
| Synopsis, 4.1.6 | Added | Added dosing schedule to be implemented in Cohort 4, based on SMC recommendation | SMC Recommendation |
| Synopsis, 3.1, 4.1.6 | Clarification | Clarified that modified induction or maintenance doses or alternative maintenance schedules may be pursued with SMC approval depending on the safety, PK and PD data observed | Informational |
| 6.1 | Clarification | Corrected typographical error | Informational |
| | | Amendment #6<br>(dated 04 January 2018) | |
| | | Revised days allowable for Cycle 1 Day 17 and Cycle | Increased flexibility at site |
| 4.2 | Revised | 2 Day 16 from ±1 day to ±2 days (Cohorts 3-7) | mercused nexionity at site |
| 4.2 | Revised | Revised days allowable for Cycle 1 Day 21 to allow +2 days (Cohorts 3-7) | Increased flexibility at site |
| 4.2 | Revised | Revised definition of "pre-dose" from within 3 hours of dosing to same calendar day of dosing (Cohorts 3-7) | Increased flexibility at site |
| 4.2 | Revised | Revised window for collection of vital signs on Cycle 1 Day and Cycle 1 Day 7 from ± 30 minutes to ± 60 minutes (Cohorts 3-7) | Increased flexibility at site |
| 4.2 | Removed | Removed vital signs and physical exam assessments on Cycle 1 Day 17 (Cohorts 3-7) | Minimize subject time at site as changes are not anticipated in specified timeframe |
| 4.2 | Deleted | Removed 4-hour post study drug administration blood hematology on Cycle 1 Days 7, 8 and 15 and removed requirement to perform pre-dose testing within 3 hours of study drug administration (Cohorts 3-7) | Minimize subject<br>discomfort as changes are<br>not anticipated in<br>specified timeframe |
| 4.2 | Deleted | Removed 4-hour post study drug administration, chemistry, coagulation, lipase, amylase & urinalysis on Cycle 1 Days 7, 8, 15 and Cycle 2 Days 8 and 15 and removed requirement to perform pre-dose testing within 3 hours of study drug administration (Cohorts 3-7) | Minimize subject<br>discomfort as changes are<br>not anticipated in<br>specified timeframe |
| 5.1 | Revised | Revised timeframe since relapse for subjects who previously received SCT (inclusion criterion #3) | Increased screening flexibility at site |
| 5.1 | Revised | Revised serum creatinine eligibility requirement (inclusion criterion #5) | Increased screening flexibility at site |
| 5.1 | Revised | Revised interval from time of previous investigational or non-investigational product treatment to start of IACS-010759 (inclusion criterion #9 and exclusion criterion #7) | Increased screening flexibility at site |
| | | Amendment #5<br>(dated 21 July 2017) | |
| Synopsis, 3.1,<br>4.1.6, 4.1.7, 7.1 | Revised | Revised the dosing regimen to include an initial Induction Phase in Cycle 1 (Day 1-7) and Maintenance Phase (Day 8-21 of Cycle 1 & Days 1-21 | PK analysis and modeling of data from cohorts 1 and 2 |

| Section | Text | Amendments | Rationale for Change |
|---|---|---|---|
| | | of all subsequent cycles) to start with subjects enrolled in Cohort 3 | |
| Synopsis | Revised | Revised the authority of the SMC to approve intermediate doses to include induction or maintenance and alternative duration of induction doses or other maintenance schedules, not to exceed 6 mg (rather than 8 mg) based on the revised dosing regimen to be initiated with subjects in Cohort 3 | Allows SMC to approve changes to the intermediate induction or maintenance doses, duration or schedules based on safety, PK & PD data without requiring a protocol amendment |
| 2.2.2 | Revised/<br>Added | Added description of results of transporter and drug-drug interaction studies | Studies complete & final data available |
| 2.2.2, 3.1, | Added | Added description of preliminary human PK data | PK analysis and modeling of data from cohorts 1 and 2 |
| 4.1.2, 4.1.7 | Revised | Revised days that PK data will be evaluated when making dose escalation decisions | Plasma concentrations will be evaluated at the end of the induction phase and again at the end of the 1 <sup>st</sup> cycle, as well as at intermediate time points, based on the revised dosing regimen |
| 4.1.7 | Clarification | Provided steady state plasma levels in ng/mL | Informational |
| 4.1.7 | Revised | Revised stopping rules to assess mean plasma concentrations at the end of the induction phase of dosing (Days 7 and 8), with additional assessments at the end of each cycle | Revised dosing regimen |
| 4.1.9 | Added | If dose interruptions occur at the end of a cycle, the new cycle will start on the first day dosing resumes | Allows appropriate collection of assessments based on study drug administration |
| 4.1.10, 4.1.11 | Deleted | Removed requirement to perform arterial blood gas (ABG) testing for all abnormal venous blood pH results | Minimize subject<br>discomfort/ will obtain for<br>DLT confirmation, where<br>needed, only |
| 4.1.11 | Added | Added anion gap calculation to be used for arterial blood collection | Informational |
| 4.2 | Added | Added new study flowchart based on revised dosing regimen to be implemented for subjects enrolled in Cohort 3-6 of the dose escalation phase and Cohort 7 of the dose expansion phase | PK analysis and modeling of data from cohorts 1 and 2 |
| 7.1 | Revised | Revised requirement for in-hospitalization from Cycle 1 Day 1 and Day 8-14 to Cycle 1 Day 7 | PK and clinical safety data from cohorts 1 and 2 |
| 8.1.3 | Deleted | Removed reference to severity grading scale for AEs not defined in the NCI CTCAE Ver 4.03 | Will assess all AEs according to CTCAE |

| Section | Text | Amendments | Rationale for Change |
|---|---|---|---|
| 8.1.3 | Added | Hospitalizations to observe subjects with elevated lactate who remain asymptomatic and would not otherwise require hospitalization will be not be considered a grade 3 toxicity for purposes of AE severity grading | Distinguishes between hospitalization being indicated due to severity of AE rather than for observation as required per protocol |
| 7.2, 7.2.1 | Clarification | Corrected typographical errors | Consistency and readability of protocol |
| | | Amendment #4<br>(dated 10 March 2017) | |
| Synopsis, 4.1.6 | Added | Added that intermediate doses of IACS-010759, not to exceed 8 mg, may also be pursued with SMC approval, depending on the safety, PK and PD data observed | Allows intermediate doses to be evaluated during the dose escalation phase based on the observed safety, PK and PD data |
| 4.1.7 | Added | Added that a cohort may be expanded to include up to 6 subjects, in the absence of a DLT in the first 3 subjects of a cohort, with SMC approval; in that instance, allocation into simultaneously enrolling cohorts will alternate between cohorts. | Recommendation by SMC during Cohort #1 review. Allows potential to further explore safety, PK and PD activity; allocation specified to reduce bias |
| 4.1.10, 4.1.11 | Clarification | Clarified that venous or arterial blood may be used to monitor lactate and blood pH; abnormal venous blood pH results will require confirmation from arterial blood. Arterial blood lactate testing will also be used to confirm a potential DLT if an abnormal venous lactate level constitutes a DLT. | Recommendation by SMC during Cohort #1 review. Not previously specified. Clarification is to ensure accuracy of lactate and blood pH results while minimizing subject discomfort, as agreed with FDA |
| 4.1.10, 4.1.11 | Revised | Revised the requirements for monitoring subjects with elevated lactate and use in DLT definition of subjects with pH between 7.30 to 7.35 who remain asymptomatic | pH results in leukemia patients can be variable and are typically lower than normal subjects. Definition revised, using recommendations from SMC during Cohort #1 review and as modified based on FDA feedback. |
| 4.1.10 | Revised | Revised the lactic acid DLT definition to include presence of clinical symptoms and specify time frame (>24 hours) to determine second episode of elevated blood lactic acid | Recommendation by SMC during Cohort #1 review. Minimum time frame added to define 2 separate episodes of elevated lactate; clinical symptoms added to reduce potential to define |

| Section | Text | Amendments | Rationale for Change |
|---|---|---|---|
| | | | a DLT based on<br>asymptomatic subjects<br>with laboratory results<br>that may be indicative of<br>disease status only, as<br>agreed with FDA |
| 4.1.15, 4.2 | Added | Additional PK and/or PD blood draws may be obtained ~every 4 days, when possible, for up to 4 weeks after last study drug administration in subjects who discontinue the study | Recommendation by SMC during Cohort #1 review. Allows potential to further explore PK and PD activity of IACS-010759 following discontinuation of study drug |
| 4.2 | Added | Additional PK blood draws on Days 8 and 14 of Cycle 2 | Allows more frequent PK<br>monitoring beyond Day<br>28, based on review of<br>available cohort 1 PK data |
| 4.2 | Added | Further additional PK blood draws during Cycle 2 at the discretion of the Principal Investigators | Allows for additional PK monitoring during Cycle 2 if needed |
| 4.2 | Added | Additional PK blood draws, weekly for the first cycle after dose-escalation | Allows monitoring of PK levels after intra-subject dose escalation |
| 4.2 | Deleted/<br>Revised | Removed Cycle 1/Day 2, Day 4, Day 9, Day 17 PD assessments and changed Cycle 1/Day 10 to also collect PD 6 hours following dosing | Revised based on review of available cohort 1 PD data |
| 5, 5.1.2, 5.2.1 | Added,<br>Clarification | Added SAS version to be used for statistical analysis; confirmed that a Statistical Analysis Plan will be prepared and finalized prior to data base lock. Clarified statistical analysis plans, including moving descriptions to different section of protocol. | Provides further information regarding planned statistical analysis; consistency and readability of protocol |
| 1, 4.1.9.2, 4.1.11 | Clarification | Corrected typographical errors | Consistency and readability of protocol |
| | | Amendment #3<br>(dated 14 December 2016) | |
| 4.1.9, 4.2 | Added | Added additional PK, lactate and blood pH testing following a dose reduction or interruption | Additional safety monitoring |
| 4.2 | Added | Added PD prior to dosing and 6 hours following dosing and PK, lactate and blood pH testing 6 hours following dosing on Cycle 1, Day 17 and Cycle 1, Day 22 | Additional safety monitoring |
| 4.1.10, 4.1.11, 4.2 | Clarification | Clarified total CO2 results will be used where bicarbonate testing is indicated | Consistency with site practice |

| Section | Text | Amendments | Rationale for Change |
|---|---|---|---|
| 4.1.11 | Revised | Updated anion gap reference range based on using total CO <sub>2</sub> results (where bicarbonate testing is indicated) | Use of total CO₂ results |
| 4.2 | Revised | ECOG testing to be performed only at Screening,<br>Day 1 of each cycle, and End of Study visits | Consistency with site practice |
| 4.2 | Clarification | Clarified coagulation testing to include INR | Inadvertently omitted in previous version |
| 4.2 | Clarification | Clarified that blood hematology results below the level of quantitation will be recorded as 0 | Informational |
| 4.2 | Clarification | Overall Response Rate assessment (as described in Section 5.2) included in study flowchart | Reminder to study personnel |
| 4.2 | Revised | Bone marrow assessments during additional cycles (beyond cycle 3) will be collected one day prior to D21 assessments | Allows bone marrow results to be available for review when performing D21 assessments |
| 4.2 | Revised | Corrected footnote 5 from 96 hours to 72 hours | Typographical error |
| | 1 | Amendment #2<br>(dated 28 October 2016) | 1 |
| 4.2, 9.1.2, 9.1.6,<br>9.1.7 | Clarification | All AEs including SAEs, should be collected, beginning from the time of the first protocol-specific intervention (study drug administration). New information regarding signs and symptoms that occurred prior to the first study medication dose on Day 1 should be recorded under the subject's Medical History. | Clarification of Adverse<br>Event Reporting |
| | | Amendment #1<br>(dated 29 August 2016) | |
| Synopsis, 4.1.6,<br>4.1.7, 7.1 | Clarification | Clarified cycle 1 length is 28 days (dosing occurs on Day 1 followed by continuous dosing starting on day 8) | FDA request |
| 4.2 | Added | Added CPK to chemistry testing | FDA request |
| 4.2 | Clarification | Clarified coagulation testing to include PT, PTT, fibrinogen | FDA request |
| 4.2 | Added | Added weekly laboratory testing during second cycle | FDA request |
| 4.1.9.2, 4.2 | Added | Added weekly laboratory monitoring during 1 <sup>st</sup> cycle of increased dose for intra-subject dose escalation | FDA request |
| 4.1.3, 6.1 | Added | Added "no available treatment options with known benefit" to subjects to be enrolled in the expansion phase | FDA request |
| 4.1.3, 6.1 | Clarification | Clarified definition of relapsed or refractory for eligibility | FDA request |
| 6.3 | Revised | Revised lactate exclusion criterion | FDA request |
| 7.2 | Added | Added description for each capsule strength | FDA request |
| 4.1.10 | Revised | Revised DLT definition | FDA request |

| Section | Text | Amendments | Rationale for Change |
|---|---|---|---|
| 4.1.11 | Revised | Revised requirements for management of elevated lactate levels, including definition of lactic acidosis symptoms | FDA request |
| 4.1.14, 4.1.7 | Clarification | Clarified PK will be evaluated in each cohort prior to dose escalation | FDA request |
| 4.1.7 | Added | Added PK levels which will pause or stop dose escalation | FDA request |
| 4.1.9 | Revised | Revised dose modification criteria to permanently discontinue study drug in any subject that develops DLT related to lactic acid | FDA request |
| 4.1.9.3 | Revised | Revised intra-subject dose escalation criteria | FDA request |
| 4.1.8 | Revised | Revised stopping rule probability statement for expansion phase | FDA request |
| 4.1.2, 4.1.7 | Added | Added safety stopping criteria to encompass toxicities beyond cycle 1 | FDA request |
| 4.1.8 | Revised | Revised the stopping boundaries for DLT monitoring to correct discrepancy | FDA request |
| 7.1 | Revised | Revised the food effect dose description to indicate the dose may be lower than R2PD | FDA request |
| 4.2 | Added | Added ECG monitoring at pre-dose and around the anticipated maximal plasma concentrations on Day 1, Day 14 and Day 28 of Cycle 1 | FDA request |
| 4.2 | Revised | Research bone marrow sample will be collected at Screening rather than Cycle 1, Day 1 | Reduce frequency of bone marrow sampling |
| 6.1 | Clarification | Revised inclusion criterion #9 to clarify the interval from prior treatment to time of initiation of study drug will be at least 2 weeks for biological/immune-based therapies | Clarification of wash-out period for prior treatment |
| 8.1 | Added | Added strong cytochrome P450 (CYP450) inhibitors or inducers as non-permitted concomitant medications | FDA request |
| 2.1 | Amended | Amended AML response rate reference | To ensure consistency with IND |
| Synopsis, 4.1.6 | Clarification | Clarified that cycles occur on a continual basis | Readability of protocol |
| 4.1.4 | Clarification | Specified number of sites | Number of sites not previously provided |
| 4.1.14 | Revised | Revised Safety Monitoring Committee representatives description to specify study-specific Medical Monitor | Responsibility transferred to CRO |
| 4.2 | Clarification | Clarified in study flow chart which study days subjects are inpatient; timing of study drug administration; cycle days | Readability of protocol |
| 4.2, 5.2 | Clarification | Clarified bone marrow aspirate/biopsy will be performed clinically as indicated, at least once per 3 cycles | To ensure consistency of testing across study subjects |
| 4.2, 10.2 | Clarification | Clarified the QTc correction formula | Informational |

| Section | Text | Amendments | Rationale for Change |
|---|---|---|---|
| 5.1.2 | Added | Added name of clinical data base to be used for study data collection | New study information |
| 7.2 | Clarification | Clarified the planned starting dose capsule strength | Informational |
| 9.1.2 | Revised | Revised clinical data base and safety data base to be used for data collection | Responsibility transferred to CRO |
| 9.1.3 | Added | Added reference to recommended AE recording guidelines | Readability of protocol |
| 9.1.7, 9.1.8 | Revised | Revised safety reporting procedures and contact information | Responsibility transferred to CRO |
| Synopsis, 4.1.7,<br>5.2.2, 6.1, 10.2 | Clarification | Corrected typographical errors | Consistency and readability of protocol |
| | | Original Protocol<br>(dated 12 April 2016) | |

## 2 Background Information

#### 2.1 AML

Acute myeloid leukemia (AML) is a malignancy of immature granulocytes or monocytes. The malignancy is characterized by accumulation of leukemic blasts and blockade of normal bone marrow production resulting in thrombocytopenia, anemia, and neutropenia. There are approximately 13,000 new cases of AML per year in the United States, with an estimated 10,000 deaths occurring in the same time period[1]. Almost all newly diagnosed cases, as well as deaths, will be in adults[2]. Standard treatment for AML includes systemic combination chemotherapy to control bone marrow and systemic disease. Treatment is generally divided into an induction phase, to attain remission, and a consolidation/maintenance phase[2].

Traditional induction chemotherapy can produce complete remissions in most (50% to 75%) subjects with AML[3, 4]. Unfortunately, between 60% and 80% of subjects with AML (especially those with adverse cytogenetic features, adverse molecular mutations or antecedent hematological disorder) will be refractory or relapse after initial response to induction therapy relapse so only 20% to 30% will achieve long-term disease-free survival. For subjects with AML refractory to initial therapy or who relapse after a brief remission (< 12 months), outcomes are more dismal. We have previously reported a median OS of 3.8 months for subjects with AML who are refractory to induction therapy [5]. Similarly subjects with relapsed AML have a poor outcome with response rates ranging from 10% to 30% and overall survival <6 months with salvage therapy[6, 7].

These results emphasize the need to explore alternate salvage regimens for subjects with relapsed/refractory AML. The development of novel and effective anti-AML agents and/or combinations is crucial to improving the outcome of AML.

Tumors frequently rewire their metabolism to ensure a steady supply of metabolites for generation of ATP and for a biosynthesis of cell constituents. While aerobic glycolysis, also known as the Warburg effect, is a common metabolic alteration in cancer, recent studies indicate that some tumors are highly dependent on oxidative phosphorylation (OXPHOS) for survival [8-13]. Several recent reports demonstrate that oxidative metabolism generates intracellular energy and metabolic intermediates necessary to promote the growth of tumor cells [14-18]. It has previously been reported that leukemia cells have increased rates of fatty acid oxidation[16] and that inhibition of fatty acid oxidation rapidly inhibits oxygen consumption and sensitizes leukemia cells to induction of apoptosis, substantiating the idea that mitochondrial oxidative metabolism supports leukemia cell survival. Another ground-breaking study has demonstrated that leukemic stem cells (LSC) are unable to utilize glycolysis when mitochondrial respiration is inhibited, indicating that the maintenance of mitochondrial function is essential for LSC survival [15]. In contrast, normal murine [19] and human hematopoietic stem cells (HSC)[15] predominantly utilize glycolysis for energy homeostasis. Therefore, inhibiting oxidative phosphorylation in the context of AML could have therapeutic potential.

#### 2.2 IACS-010579

#### 2.2.1 IACS-010759 Preclinical Biology

IACS-010759 inhibits complex I of mitochondria oxidative phosphorylation (OXPHOS). IACS-010759 is a potent inhibitor of the proliferation of human cancer cells, including AML cell lines, human primary AML cells, and glycolysis-deficient NB-1 neuroblastoma cells. Both primary AML


cells and established cell lines demonstrated dose-dependent growth inhibition and reduction of cell viability in response to IACS-010759, with IC $_{50}$  values ranging from 1-10 nM. Ectopic expression of the yeast complex I protein NDI-1 partially restored AML cell viability, indicating that the effects of IACS-010759 were mechanism-based *via* OXPHOS inhibition. In contrast to the potent effect of IACS-010759 on the viability of tumor cells, the compound had minimal effects on the viability of bone marrow cells obtained from healthy subjects, suggesting that the compound has a therapeutic window for tumor cells *vs.* normal leukocytes.

The sensitivity of NB-1 cells, which lack the gene that encodes the essential glycolytic pathway enzyme phosphogluconate dehydrogenase (PGD), to IACS-010759 was reduced upon ectopic expression of PGD. This suggests that the sensitivity of NB-1 cells to IACS-010759 is due to their inability to upregulate glycolysis in response to energy stress conferred by IACS-010759 treatment. This is consistent with the OXPHOS inhibitory mechanism of IACS-010759 and with the observed increase in potency of IACS-010759 to kill AML cells compared to normal bone marrow cells.

IACS-010759 inhibits tumor growth and extends survival in AML xenograft models. IACS-010759 caused dose-dependent tumor regression or substantial tumor growth inhibition (TGI) in both orthotopic and subcutaneous xenograft models with human AML and NB-1 neuroblastoma cells, while overall survival was increased in both primary AML and OCI-AML3 cell line orthotopic xenograft models.

In these *in vivo* efficacy experiments, increases in dose or shortening of the dosing interval corresponded to increases in efficacy, measured as TGI or regressions. Notably, in all studies, decreases in dosing frequency at a given dose correspond to decreases in efficacy, with QD dosing being more effective than intermittent dosing of the same dose of IACS-010759.

Trough plasma levels at steady state of 10-20 nM (5.6-11.3 ng/mL) were associated with efficacy in these xenograft studies, regardless of the dosing regimen. This concentration correlates well with the IACS-010759 concentrations of 1-10 nM that are required to inhibit cancer cell proliferation and to inhibit the OXPHOS pathway in cell based assays *in vitro*. Based on these preclinical efficacy studies, it seems reasonable to target sustained trough steady state plasma levels of 10-20 nM (5.6-11.3 ng/mL) IACS-010759 for efficacy in human clinical trials.

#### 2.2.2 IACS-010759 Nonclinical Experience

The pharmacological, pharmacokinetic, and toxicological properties of IACS-010759 were characterized in a series of completed and ongoing nonclinical studies. These studies demonstrate that:

- IACS-010759 inhibits proliferation and reduces the viability of primary human AML samples treated *ex vivo* and in AML cell lines with IC₅₀ values ranging from 1-10 nM, and has minimal effects on the viability of bone marrow cells obtained from healthy subjects. These studies suggest that IACS-010759 has a therapeutic window for tumor cells vs. normal leukocytes.
- IACS-010759 caused dose-dependent tumor regression or substantial tumor growth inhibition (TGI) in both orthotopic and subcutaneous xenograft models with human AML and NB-1 neuroblastoma cells. In addition, survival was increased in both primary AML and OCI-AML3 cell line orthotopic xenograft models. Several oral dosing regimens were explored in these studies, and efficacy was consistently observed with steady state trough plasma levels of 10-20 nM (5.6-11.3 ng/mL) IACS-010759.

- IACS-010759 had negligible inhibitory activity (estimated IC<sub>50</sub> > 30  $\mu$ M) at hERG K<sup>+</sup> channels and did not prolong the QTc interval in monkeys at doses up to 1.5 mg/kg/day for up to 28 days.
- IACS-010759 did not elicit central nervous system effects in rats treated with oral doses up to 2 mg/kg based on neurobehavioral parameters (functional observation battery).
- IACS-010759 exhibited low plasma clearance, a high volume of distribution, and a long half-life (42 to 57 hours) in mice, rats, dogs, and monkeys. Upon oral dosing, the compound was absorbed relatively slowly, with Tmax values in the range of 3 to 8 hours and bioavailability of ~100% in mouse and rat and ~36% in monkey.
- IACS-010759 exhibited low/moderate metabolic turnover following incubation with liver microsomes and hepatocyte preparations from mouse, rat, dog, monkey and human. No metabolites unique to human were identified. IACS-010759 was found to be a moderate competitive inhibitor of CYP 2C19 (IC<sub>50</sub> = 4 uM), but did not inhibit any other CYP isoforms tested. No time dependent inhibition of CYPs 1A2 or 3A4 was observed.
- The potential for CYP enzyme induction by IACS-010759 could not be assessed in standard hepatocyte enzyme induction assays, likely because of the mechanism-based effects of IACS-010759 on oxidative phosphorylation. Therefore, the potential of IACS-010759 to reduce the levels of drugs metabolized by CYP450 enzymatic pathways is unknown.
- In transporter studies, IACS-010759 had no effect on BSEP-, MDR1-, OAT1-, OAT3-, OATP1B1-, OATP1B3- and OTC1-mediated probe substrate transport. IACS-010759 moderately inhibited the BCRP- and OCT-2 mediated probe transport by 27% and 36%, respectively, at 1  $\mu$ M. IACS-010759 is likely a substrate of the BCRP and MDR1 transporters.
- A drug-drug interaction (DDI) study was conducted with IACS-010759 and pentagastrin or the histamine H2 blocker famotidine in dogs. Neither pentagastrin nor famotidine affected the plasma levels of IACS-010759 after oral administration, indicating low potential for DDI with drugs that affect stomach pH.
- IACS-010759 was nongenotoxic in a bacterial reverse mutation assay without or with metabolic activation, and in a bone marrow micronucleus test conducted after 28-days of oral administration in rats at doses up to 2 mg/kg/day, the highest dose tested.
- Single-dose IV administration of IACS-010759 to monkeys showed that sporadic emesis observed following oral and IV administration was a systemic rather than a local GI effect. Plasma levels of IACS-010759 associated with acute emesis were higher than those not associated with emesis.
- IACS-010759 was well tolerated in GLP-compliant 28-day oral toxicity studies in rats and monkeys at doses up to 1 mg/kg/day and 1.5 mg/kg/day, respectively. Higher doses in the 28-day studies and/or 14-day dose range-finding studies resulted in adverse effects in both species, including moribundity requiring euthanasia and/or mortality in rats at ≥2 mg/kg/day and in monkeys at ≥3 mg/kg/day. There were no treatment-related histopathological findings in tissue sections from the 28-day studies.
- C<sub>max</sub> on Day 28 from pivotal toxicity studies was 61.3 ng/mL in rats and 99.3 ng/mL in monkeys at doses of 1 mg/kg/day and 1.5 mg/kg/day, respectively. These C<sub>max</sub> values, which were observed at doses that were well tolerated for 28 days in each species, were notably higher than steady state trough plasma levels of 5.6 11.3 ng/mL at which efficacy was consistently observed in nonclinical xenograft models of human tumor cells. Because the human peak:trough plasma levels with daily oral dosing are projected to be <2-fold based on projected human clearance and on the preliminary data from cohorts 1 and 2 of the</p>

present study, this represents a significant exposure multiple above the projected human exposure required for efficacy.

#### 2.2.3 IACS-010759 Chemical Properties

IACS-010759 is available as a crystalline hydrochloride salt, with the chemical name 5-(5-methyl-1-(3-(4-(methylsulfonyl)piperidin-1-yl)benzyl)-1H-1,2,4-triazol-3-yl)-3-(4-(trifluoromethoxy)phenyl)-1,2,4-oxadiazole hydrochloride salt.

The molecular formula of IACS-010759 hydrochloride salt is  $C_{25}H_{25}F_3N_6O_4S$ .HCl and the molecular weight is 599.024 g/mole (562.564 g/mole as the free base). This compound has not yet been assigned a generic name.

## 3 Study Rationale

#### 3.1 Rationale for IACS-010759 Dose Selection

The starting dose of IACS-010759 has been selected as the human equivalent dose corresponding to no more than 1/10 the no observed adverse effect level (NOAEL) in nonclinical toxicology studies. Additional considerations for dose selection include avoiding C<sub>max</sub>-associated emesis and anticipation of achieving plasma levels associated with preclinical efficacy within a reasonable number of escalation steps. IACS-010759 was well tolerated in 28-day oral toxicology studies in the monkey and rat and the NOAEL in those studies were 1.5 mg/kg/day and 1 mg/kg/day, respectively. Based on these considerations, our projection is that a human starting dose of 0.5 mg will allow a thorough exploration of safety and tolerability in humans while minimizing the exposure of subjects to doses not anticipated to be effective. Using a model based on allometric scaling, a human dose of 0.5 mg, given once daily, would be anticipated to produce a C<sub>max</sub> of ~2.3 ng/mL and to give a projected steady state exposure ratio, animal-tohuman, of approximately 27-fold based on the 1 mg/kg/day dose in the rat and 43-fold based on the 1.5 mg/kg/day dose in the monkey for C<sub>max</sub> and approximately 7-fold based on the rat and 11-fold based on the monkey for AUC. Therefore, the human starting dose of 0.5 mg of IACS-010759, administered orally once daily, would be anticipated to be safe and well tolerated, while allowing attainment early in the dose-escalation studies of doses that may be projected to show benefit in patients.

Limited PK data from subjects in cohorts 1 and 2 showed unexpected levels of accumulation of IACS-010759 throughout the dosing period, consistent with a model in which the clearance of IACS-010759 decreases exponentially with time, leading to an increasingly long terminal  $T_{1/2}$  and accumulation upon multiple dosing. A mathematical model and simulation has been developed based on data from the subjects treated with IACS-010759 to date that predicts the observed human PK. Based on this model, a modified dosing regimen is being implemented for the dose escalation phase with cohorts 3-6 and for the dose expansion phase with cohort 7, consisting of an induction phase in which IACS-010759 is administered daily for up to 7 days, followed by a maintenance phase in which a lower dose is administered weekly to maintain steady state plasma levels (or as otherwise specified by the SMC based on safety, PK and PD data observed).


### 3.2 Rationale for Study Design

Current treatment options for relapsed or refractory AML reflect an unmet medical need and additional options for treatment are needed.

Preclinical data reviewed above strongly suggest a robust antitumor activity with IACS-010759 in AML. The current study focuses on evaluating the maximum tolerated dose (MTD), recommended phase 2 dose (RP2D) and safety profile of IACS-010759 and preliminary clinical efficacy in subjects with confirmed relapsed or refractory AML and no available treatment options with known benefit.

The results from this study will form the basis for decisions for future studies.

## 4 Experimental Plan

## 4.1 Study Design

#### 4.1.1 Study Phase

Phase 1 study with a dose-escalation phase followed by an expansion phase.

#### 4.1.2 Enrollment/Randomization

This open label study will employ a sequential-cohort, non-randomized, single site enrollment. The study will be under ongoing review by a Safety Monitoring Committee (see section 4.1.14).

In the dose-escalation phase, all subjects in a cohort will be monitored for DLT for the first cycle before proceeding with subsequent cohorts. To assess toxicities that may occur beyond cycle 1, cohorts of up to 6 subjects will be assessed following completion of 4 cycles of study drug. If two or more subjects in the cohort did not receive at least 80% of the planned dose due to adverse events, dose escalation will be paused and an evaluation will be performed.

#### 4.1.3 Subject Population

For complete subject eligibility please see section 5.

Dose-escalation phase: Subjects with confirmed relapsed or refractory AML and no available treatment options with known benefit.

Expansion phase: Subjects with relapsed or refractory AML who have failed therapy with up to one prior salvage regimen and no available treatment options with known benefit.

Exception: stem cell transplant [SCT] or stem cell therapy for subjects who previously underwent SCT/stem cell therapy, and are currently in remission will not be considered a salvage regimen.

Relapsed or refractory status is defined by the failure of at least one prior cycle of chemotherapy (including but not limited to cytotoxic chemotherapy, hypomethylator therapy, immune-based therapy, stem cell transplant or stem cell therapy, FLT3-inhibitor therapy, investigational therapy, and others). Patients in first relapse and less than 12 months from diagnosis [short first remission] or in second or later relapse are eligible.


#### 4.1.4 Number of Sites and Subjects

2 to up to 48 subjects will be enrolled at one site.

#### 4.1.5 Sample Size Considerations

The dose-escalation phase of the study will enroll 3-6 subjects in each cohort, based on a 3+3 dose-escalation design to assess the MTD level. A maximum of 36 subjects will enroll in the dose-escalation phase.

A maximum of 18 subjects will enroll in the expansion phase (12 additional subjects and the 6 subjects from the dose-escalation phase at the cohort of the highest dose level shown to be well tolerated or the RP2D). The expansion phase sample size of 18 subjects is not based on a formal sample size calculation. Rather, 18 subjects are deemed to be sufficient for the assessment of safety and tolerability as the primary objective and the exploration of clinical anti-tumor activity and other secondary and exploratory endpoints.

#### 4.1.6 Treatment Cohorts and Treatment Schema

In cohorts 1 and 2, IACS-010759 was administered orally daily on a continual 21-day schedule (1 cycle = 21 days of daily dosing), with the exception that the first cycle for each subject contains a 7-day single dose lead-in (first cycle = 28 days). Starting on day 8 of cycle 1 for subjects enrolled in cohorts 1 and 2, dosing is on a 21 day schedule until confirmed PD, initiation of alternative cancer therapy, unacceptable toxicity, or other reasons to discontinue treatment prematurely occur as defined in Section 4.1.9.

Based on PK modeling of data from cohorts 1 and 2, the dose regimen for cohort 3 and subsequent cohorts will change to include an induction phase with daily dosing, followed by a maintenance phase at a dose sufficient to maintain the steady state levels achieved during the induction phase. In these cohorts, IACS-010759 will be administered orally daily (up to 7 days) during the induction phase(Cycle 1, Days 1-7). Starting on day 8 of cycle 1 for all cohorts, maintenance dosing will be administered on a 21-day schedule until confirmed PD, initiation of alternative cancer therapy, unacceptable toxicity, or other reasons to discontinue treatment prematurely occur as defined in Section 4.1.9.

The planned dose levels are given in Table 1 and 2, below:

Table 1: Dosing schema for Cohorts 1 and 2

| PHASE | COHORT | NO OF SUBJECTS | IACS-010759 DOSE LEVEL * |
|------------|----------|----------------|--------------------------|
| Dose- | Cohort 1 | 3-6 | 0.5 mg |
| escalation | Cohort 2 | 3-6 | 1 mg |

<sup>\*</sup>Intermediate doses of IACS-010759, not to exceed 8 mg, not listed above may also be pursued with SMC approval, depending on the safety, PK and PD data observed.

Table 2: Revised dosing schema for Cohorts 3-6 (Dose-Escalation) and Cohort 7 (Dose Expansion)

| PHASE | COHORT | NO OF<br>SUBJECTS | INDUCTION DOSE*<br>(FREQUENCY#) | MAINTENANCE DOSE*<br>(FREQUENCY#) |
|---|---|---|---|---|
| | Cohort 3 | 3-6 | 2 mg (daily, Cycle 1 Day 1-7) | 0.5 mg (once per week) |
| Dose- | Cohort 4** | 3-6 | 2.5 mg (daily, Cycle 1 Day 1-7) | 1.0 mg (three times per week) |
| escalation | Cohort 5 | 3-6 | 2.5 mg (daily, Cycle 1 Day 1-5) | 1.5 mg (three times per week) |
| | Cohort 6 | 3-6 | 3 mg (daily, Cycle 1 Day 1-5) | 2 mg (three times per week) |
| Expansion | Cohort 7 | 12 | RP2D | RP2D |

<sup>\*</sup>Intermediate induction or maintenance doses of IACS-010759 may be pursued with SMC approval, not to exceed 6 mg, and

<sup>#</sup> alternative duration of induction doses or other maintenance schedules not listed above may also be pursued with SMC approval depending on the safety, PK and PD data observed.

<sup>\*\*</sup>Following their review of Cohort 3, the SMC recommended implementation of the following dose schedule for

subjects who enroll in Cohort 4 of the study:

Induction dose: 2.5 mg, administered daily, Cycle 1 Day 1 through Day 7

Maintenance dose: 1 mg, administered 3x/week (for a total weekly dose of 3 mg) with the first maintenance dose starting on Cycle 1 Day 8

#### 4.1.7 Dose-escalation

A standard 3+3 dose-escalation design will be used to determine MTD. The potential dose schedule is shown in section 4.1.6. In the first cohort, as a safety precaution, each new subject began treatment only after the safety analysis for DLTs and evaluation of PK data during the first cycle (28 days) was completed for the previous subject. In subsequent cohorts of the dose-escalation phase, new subjects will be entered and treated only after the previous subject has been treated with IACS-010759 for up to 7 days (e.g., has completed the induction phase) and DLT safety analysis for each subject will be performed after completion of cycle 1. PK data will be monitored for each subject and evaluated for each cohort during the study and plasma levels will be considered when making dose escalation decisions.

The following dose-escalation rules will be applied:

- If 0 out of the 3 subjects have a DLT, the next cohort may be started.
- If 1 out of the 3 subjects has a DLT, an additional 3 subjects will be enrolled in the same cohort. If none of these 3 additional subjects have a DLT after being observed for 28 days (i.e., cycle 1), the next dose escalation cohort may be started.
- If 2 or more out of 6 subjects in Cohort 1 develop a DLT, enrollment will cease immediately and the study will be halted. No MTD can be determined.
- If 2 or more out of 6 subjects in the following Cohorts (2-6) develop a DLT, enrollment into the cohort will cease, and the prior cohort's dose level will be deemed as MTD level. All subjects from the non-tolerated cohort will be de-escalated to the prior cohort's dose level.
  - If at least 2 of 3 or 2 of up to 6 patients experience a DLT at a given dose, then the MTD has been exceeded (stopping dose). Once the MTD has been exceeded, treat another 3 patients at the previous dose if there were only 3 patients treated at that dose.

During dose escalation, if necessary, cohorts may be expanded in the absence of a DLT, to a total of up to 6 subjects to further explore safety, PK and PD activity of IACS-010759 at each dose level with the approval of the SMC. Such an expansion may occur concurrently with dose escalation to the next dose level. A predetermined allocation to cohorts that minimizes selection bias will be used when enrolling into two open cohorts simultaneously. Allocation to simultaneously open cohorts will be performed in an alternating random manner, based on entry into the study. During dose escalation, intermediate (including induction or maintenance) doses and alternative duration of induction doses or other maintenance schedules of IACS-010759, not to exceed 6 mg, may also be pursued with SMC approval, depending on the safety, PK and PD data observed.

The dose escalation phase of the study will be paused after the dose at which the mean steady state plasma levels, measured as pre-dose concentrations on Day 28 for cohorts 1 and 2 and as pre-dose concentrations on Day 8 (e.g. the end of the induction phase) for cohorts 3 onwards, reach levels of  $\geq$ 20 nM (11 ng/mL). A full review of the safety, PK and efficacy data from that

cohort will be performed and escalation may be continued if the MTD has not been reached, and the Sponsor obtains agreement with FDA to continue dose escalation.

The dose escalation phase of the study will stop after the dose for which the mean Cmax on Day 28 for cohorts 1-2 or Day 7 for cohorts 3 and onwards is  $\geq$ 100 nM, or after the dose for which the mean steady state concentration for the cohort, as measured on the last day of any 21 day Cycle, is  $\geq$ 100 nM, whichever dose is lower.

To assess toxicities that may occur beyond cycle 1, cohorts of up to 6 subjects will be assessed following completion of 4 cycles of study drug. If two or more subjects in the cohort did not receive at least 80% of the planned dose due to adverse events, dose escalation will be paused and an evaluation will be performed.

Once the MTD has been established or the dose-escalation completed without identifying a MTD, the RP2D will be defined based on an assessment the safety, pharmacokinetic (PK), pharmacodynamic (PD), biomarker, and response data.

At the discretion of the sponsor, dose-escalation may be stopped before an MTD is reached. In this case, the RP2D may be chosen based on an assessment of the safety, PK, PD, biomarker, and response data evaluable up to that time. An MTD does not have to be reached to expand a dose cohort if the available data demonstrate that a lower dose level may provide antitumor activity while minimizing potential risk. Upon completion of the dose-escalation, the cohort with either the highest dose level shown to be well tolerated or the RP2D will be expanded to a total of 6 subjects (if not already expanded to 6 subjects due to either observation of a DLT or to further explore safety, PK and PD activity of IACS-010759 at that dose level).

Late onset DLTs that could not be taken into consideration prior to scheduled dose escalations will be ad-hoc evaluated on a case-by-case basis, and may lead to enrollment of additional subjects in specific cohorts or to revision of the previously determined MTD.

#### 4.1.8 Expansion Phase

Subjects in the expansion phase will be treated at the RP2D level determined in the dose-escalation phase.

The primary objective of the expansion phase is to determine safety of IACS-010759.

Additionally, as part of the expansion phase, the effect of a high fat meal on the PK of IACS-010759 (Food Effect) will be evaluated in a total of 6 subjects (Food Effect cohort), as described in Section 7.1. After the first 6 subjects have been enrolled in the expansion cohort, the next 6 subjects will be enrolled in the Food Effect cohort.

To evaluate safety, the method of Thall, Simon and Estey [20] will be used for monitoring DLTs occurring in the first cycle. The probability of DLT is denoted by  $P_T$ . We assume  $P_T \sim$  beta (0.4, 1.6). Our stopping rule is given by the following probability statement:  $Pr(P_T > 0.20 \mid data) > 0.80$ .

That is, if at any time during the study we determine that there is more than 80% chance that the unacceptable toxicity rate is more than 20% during the expansion phase, then the enrollment will be stopped. Subjects will be monitored by a cohort size of 6 during the expansion phase according to the following stopping boundaries for DLTs, starting from the 12th

subject. The monitoring rule for DLTs, based on these assumptions and monitoring conditions is found in Table 3. For example, accrual in the expansion phase will cease if 4 or more subjects experience DLTs among the first 12 subjects. The operating characteristics are summarized in Table 4. The design software Multc Lean Desktop (version 2.1) developed by the Department of Biostatistics at M. D. Anderson Cancer Center was used to generate the toxicity stopping boundaries and the operating characteristics tables.

Table 3 Stopping boundaries for DLT monitoring

| # Subjects evaluated | 12 | 18 |
|----------------------|------|------|
| # Subjects with DLTs | 4-12 | 6-18 |

Table 4 Operating characteristics of toxicity monitoring

| True DLT Rate | Early Stopping Probability | Average Sample Size |
|---------------|----------------------------|---------------------|
| 0.10 | 0.0256 | 17.8 |
| 0.15 | 0.0922 | 17.4 |
| 0.20 | 0.2054 | 16.8 |
| 0.25 | 0.3512 | 15.9 |
| 0.30 | 0.5075 | 15.0 |

#### 4.1.9 Dosing Adjustments, Delays and Discontinuations

IACS-010759 dose reduction/interruption/discontinuation decisions should be based on the CTCAE version 4.03 of the toxicity and according to the guidelines shown below. If toxicity is not covered in the table, doses may be reduced or held at the discretion of the investigator for the subject's safety. Additional PK, blood pH and lactate testing will be performed following a dose reduction or resumption of dosing following a dose interruption, as described in Section 4.2. IACS-010759 should be permanently discontinued in any subject that develops DLT due to lactic acid.

If a dose interruption occurs at the end of a cycle, the next cycle will be delayed and start on the first day of dosing of the next cycle. Dose interruptions which occur during a cycle will not change the study days during the cycle.

#### 4.1.9.1 IACS-010759 Dose Adjustments for Drug-Related Hematological AEs

- Subjects with acute leukemias usually present with abnormal peripheral blood counts at the
  time therapy is started and myelosuppression is an expected event during the course of
  therapy for acute leukemias. Thus, no dose adjustments or treatment interruptions for
  myelosuppression will be planned for the first 4 cycles and/or in the presence of residual
  leukemia. After that, treatment interruptions and dose adjustments may be considered
  according to the following guidelines only when there is no evidence of residual leukemia.
- Subjects with a response (e.g., no evidence of residual leukemia or cytopenias not considered to be related to leukemia) and pre-cycle counts of neutrophils >1.0 x  $10^9$ /L and platelets >50 x  $10^9$ /L who have sustained low counts of neutrophils <0.5 x  $10^9$ /L or a platelet count <20 x  $10^9$ /L for more than 2 consecutive weeks in the current cycle, may have the treatment with IACS-010759 interrupted at the discretion of the treating physician after discussing with the Principal Investigator (PI) until neutrophils recover to  $\ge 0.5 \times 10^9$ /L and platelets to  $\ge 30 \times 10^9$ /L. If prolonged myelosuppression defined as ANC <  $0.5 \times 10^9$ /L and

platelets  $< 20 \times 10^9$ /L (more than 6 weeks) with evidence of a hypocellular marrow (marrow cellularity less than 5% without evidence of leukemia) is observed, IACS-010759 will be discontinued in these subjects. Delays in the start of subsequent cycles greater than 6 weeks will be acceptable only for subjects who are deriving clinical benefit and after discussion with the Principal Investigator (PI) of potential risk/benefit ratio and complete documentation of the degree of clinical benefit and reason for continuation on this regimen.

- If there are persistent peripheral blood blasts, or the bone marrow shows >5% blasts or evidence of leukemia, treatment may be continued regardless of neutrophil and platelet count with supportive care as needed. Dose-interruptions of IACS-010759 in these subjects should be considered on an individual case and discussed with the PI and the sponsor.
- Subjects with a response (no marrow evidence of leukemia) and pre-cycle counts of neutrophils <1x10<sup>9</sup>/L and platelets <50 x10<sup>9</sup>/L may be continued regardless of neutrophil and platelet count with supportive care as needed. Dose-interruptions in these subjects should be considered on an individual case and discussed with the PI and the sponsor.

4.1.9.2 IACS-010759 Dose adjustments for Non-Hematologic Drug-Related AEs Dose adjustments for AEs will be performed using dose levels suggested in Table 1 and 2 in Section 4.1.6. Thus, if cohort 6 is established as the MTD, one and two dose level reductions of IACS-010759 will be the doses specified in cohort 5 and cohort 4, respectively. If the MTD is below cohort 3 further dose reduction levels of IACS-010759 will be defined before moving to the expansion phase of the study to allow for the below specified dose-reductions.

Table 5: Dose adjustments for non-hematologic drug-related AEs, clinically significant in the opinion of the investigator

| Grade | Occurrence | Dose modification |
|---|---|---|
| 1 or 2 | Any time | No dose reduction. |
| (Persistent grade 2: Consider similar dose adjustments if persistent and not | 1st and 2nd<br>time | Hold treatment with IACS-010759. Resume IACS-010759 at pre-interruption dose if recovery to ≤ Grade 1 or baseline occurs within 14 days. If toxicity persists for >14 days, hold therapy and resume at ONE dose level below current dose for IACS-010759 ONLY after recovery of toxicity to ≤ Grade 2. Dose re-escalation to prior dose of IACS-010759 is not permitted. |
| responding to optimal management in the opinion of PI and treating physician) | 3rd time | Stop treatment with IACS-010759 and discontinue subject. (For subjects with clinical benefit/response from IACS-010759 we will consider continuation if toxicities resolve to ≤ grade 1 and with proper dose adjustments after consultation with the PI and the sponsor) |
| 4 | Any time | Stop treatment with IACS-010759 and discontinue subject. (For subjects with clinical benefit/response from IACS-010759 we will consider continuation if toxicities resolve to ≤ grade 1 and with proper dose adjustments after consultation with the PI and the sponsor) |

These general guidelines constitute guidance to the Investigator and may be supplemented by discussions with the Medical Monitor representing the Sponsor in specific cases.

#### 4.1.9.3 *Intra-Subject Dose Escalation*

Intra-subject dose escalation of IACS-010759 (in accordance with the dosing schema in Table 1 and 2) will be permitted provided:

- Subject has completed ≥2 cycles at their current dose level and has not achieved a CR or Cri
- Subject has not experienced any grade 3 or higher non-hematologic drug-related toxicity, and

Subject has not experienced DLT,

- The dose may be escalated by one dose level no more frequently than every 2 cycles.
- The escalated dose level must have been fully evaluated and shown not to exceed the MTD (0 DLT of 3 or ≤1 DLT of 6)

If an intra-subject dose escalation occurs, laboratory monitoring will be increased to weekly during the first cycle of the increase dose.

#### 4.1.9.4 Other Allowable Modifications of Dose Schedules

Other modifications of dose schedules than the above will be allowed within the following guidelines:

- Further dose reductions can be made to keep clinically significant toxicities grade < 2.
   <p>Dose adjustments by more than 1 dose level at a time (e.g., from cohort 6 dose to cohort 4 dose) can be considered when judged in the best interest of the subject (e.g. severe myelosuppression, lactic acidosis) when the toxicity has resolved. The reason for this reduction will be discussed with the PI or Co-PI and documented in the medical record.
- Treatment interruptions and dose modifications other than the ones mentioned above can be considered after discussion with the PI, sponsor and proper documentation of the rationale.

#### 4.1.10 DLT, MTD and RP2D definitions

The MTD is defined as the highest dose studied for which the observed incidence of DLT is less than 33%. Frequencies of toxicities will be tabulated according to the NCI Common Toxicity Criteria version 4.03.

The RP2D will be determined based on the safety data and all available correlative data from the escalation phase by the Safety Monitoring Committee.

Dose-limiting toxicity (DLT) is defined as a clinically significant non-hematologic adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications and is possibly, probably or definitely related to the study drug and occurring during the first cycle (21 days) on study that meets any of the following criteria:

- All Grade 4 non-hematologic toxicities of any duration
- All grade 3 non-hematologic toxicities. Exceptions are as follow:
  - Grade 3 nausea, vomiting and diarrhea that does not require hospitalization or TPN support and can be managed with supportive care to ≤ grade 2 within 48 hours.
  - Grade 3 electrolyte abnormalities that are corrected to ≤ grade 2 within 24 hours

#### Lactic Acid:

- Blood lactic acid levels [>4.0 mmol/L]) and decreased blood pH (>7.2 to <7.30) and no clinical symptoms of metabolic acidosis [nausea, vomiting, generalized muscle weakness, tachycardia, hypotension and rapid breathing] and normal potassium maintained in two consecutive laboratory assessments separated by >12 hours despite management as described in Section 4.1.11. To qualify as a DLT, the blood lactic acid levels [>4.0 mmol/L]) and decreased blood pH (<7.30) should be confirmed on arterial blood draws. Patients who develop pH between 7.30 - 7.35 while on therapy who are asymptomatic, and have other etiologies for metabolic acidosis ruled out, may be permitted to continue on treatment. These patients will have an increased monitoring of pH and lactate levels minimally at approximately 6 hours, 12 hours and 24 hours, until normalization of pH is established, so as to rule out any worsening acidosis. Patients with a baseline normal pH (>7.35) and no clinical evidence of progressive leukemia (defined by >50% blasts in the bone marrow or peripheral blood, white count >20K, requiring hydroxyurea to control WBC counts, or new extramedullary leukemia) who develop acidosis that fulfills the criteria for a DLT during the DLT window, should be considered a DLT.
- Blood lactic acid levels [>4.0 mmol/L]), decreased blood pH (<7.35 if the</li>

baseline pre-therapy pH was >7.35 or blood pH <7.30 if the baseline pre-therapy pH was  $\leq$ 7.35), with bicarbonate >LLN and anion gap elevated, abnormal potassium and/or, in the opinion of the investigator, the subject is symptomatic for lactic acidosis [nausea, vomiting, generalized muscle weakness, tachycardia, hypotension and rapid breathing (Section 4.1.11, point 3). To qualify as a DLT, the blood lactic acid levels [>4.0 mmol/L]) and decreased blood pH <7.35 if the baseline pre-therapy pH was >7.35 or blood pH <7.30 if the baseline pre-therapy pH was  $\leq$ 7.35), should be confirmed on arterial blood draws.

 Second episode of blood lactic acid level > 4.0 mmol/L, confirmed as lactic acid level > 4.0 mmol/L on arterial blood, separated by >24 hours blood draw, in the presence of clinical symptoms attributable to lactic acidosis [nausea, vomiting, generalized muscle weakness, tachycardia, hypotension and rapid breathing]

Myelosuppression and associated complication are expected events during leukemia therapy. Only prolonged myelosuppression, as defined as ANC <500 through day 42 or later (6 weeks) from start of therapy without any evidence of leukemia, will be considered in defining the MTD and DLT.

#### 4.1.11 Assessment of Elevated Lactic Acid Levels

Lactic acidosis is a potential mechanism-based side effect resulting from inhibition of mitochondrial oxidative phosphorylation by IACS-010759 and has been observed at high doses in preclinical studies. Peripheral venous or arterial lactate levels will be monitored during the trial as detailed in section 4.2 study flowchart. (Note: Venous or arterial blood may be used to monitor lactate and blood pH. Arterial blood lactate testing will also be used to confirm a potential DLT if an abnormal venous lactate level constitutes a DLT.)

A recent review by Kruse et al. [21] on the measurement of lactate concluded that peripheral venous lactate levels are highly correlated with arterial blood lactate levels. In the setting of elevated lactate, a complete physical exam and directed history will be performed to rule out other causes of elevated lactate levels (see appendix 9.1)

Subjects will have their lactic acid levels, blood pH as well as electrolytes including chloride and bicarbonate (reported as total CO<sub>2</sub>) levels measured according to section 4.2. Subjects with lactate levels >4 mmol/L and pH <7.30 and symptoms attributable to lactic acidosis [nausea, vomiting, generalized muscle weakness, tachycardia, hypotension and rapid breathing] will be hospitalized for monitoring of lactate levels and pH, electrolytes and symptoms of lactic acidosis [nausea, vomiting, generalized muscle weakness, tachycardia, hypotension and rapid breathing] for a minimum of 24 hours. The lactic acid and blood pH levels will be assessed as follows:

1. If lactic acid is > ULN but below 4.0 mmol/L, pH >7.35 and subject is asymptomatic, treatment can be continued. Patients with pH between 7.30 - 7.35 who are asymptomatic, and have other etiologies for metabolic acidosis ruled out, may be permitted to continue on treatment. These patients will have an increased monitoring of pH and lactate levels minimally at 6 hours, 12 hours and 24 hours, until normalization of pH is established, so as to rule out any worsening acidosis. Patients with a baseline normal pH (>7.35) and no clinical evidence of progressive leukemia (defined by >50% blasts in the bone marrow or peripheral blood, white count >20K, requiring hydroxyurea to control WBC counts, or new extramedullary leukemia) who develop acidosis that fulfills the criteria for a DLT during the DLT window, should be considered a DLT.

- 2. If lactic acid >ULN but below 4.0 mmol/L, and subject is symptomatic (nausea, vomiting, generalized muscle weakness, tachycardia, hypotension and rapid breathing), treatment should be interrupted as indicated and lactic acidosis workup performed.
- 3. If lactic acid is above 4.0 mmol/L, blood pH ≥7.35 and bicarbonate (reported as total CO<sub>2</sub>) is <LLN, potassium is normal and anion gap <14, and subject is asymptomatic, dosing should be interrupted. Lactic acid and blood pH and electrolytes should be reassessed within 12 hours on arterial and/or venous blood draw until the lactic acid level is <4.0 mmol/L. Once the lactic acid level is <4.0 mmol/L on arterial and/or venous draw, the subject can continue therapy at the discretion of the investigator.
- 4. If lactic acid is above 4.0 mmol/L, blood pH <7.35 if the baseline pre-therapy pH was >7.35 or blood pH <7.30 if the baseline pre-therapy pH was ≤7.35) and the bicarbonate (reported as total CO₂) is <LLN and anion gap is elevated, and/or the subject is symptomatic, this will be considered a DLT. Treatment should be interrupted and lactic acidosis workup performed (See Section 7.2.3).</p>

Anion gap via venous blood collection can be calculated as follows: Anion Gap= [Na+] - [Cl-] - [total CO<sub>2</sub>]; normal range 4-14 mmol/L.

Anion gap via arterial blood collection can be calculated as follows: Anion Gap= [Na+] - [Cl-] - [HCO3-]; normal range 8-16 mEq/L.

Symptoms of lactic acidosis include nausea, vomiting, generalized muscle weakness, tachycardia, hypotension and rapid breathing. Subjects with clinical symptoms concerning for lactic acidosis should have an arterial blood gas assessment. Lactic acidosis is characterized by an elevated blood lactate concentration [>4.0 mmol/L]), decreased blood pH (<7.35), and electrolyte disturbances with an increased anion gap.

#### 4.1.12 Subject Withdrawal

In the absence of treatment delays due to adverse events, treatment may continue until one of the following criteria applies:

- 1. Clinically significant progressive disease, or
- 2. Intercurrent illness that prevents further administration of treatment, or
- 3. Subject request, or
- 4. General or specific changes in the subject's condition render the subject unacceptable for further treatment in the judgment of the investigator, or
- 5. Unacceptable toxicity that in the opinion of the investigator makes it unsafe to continue therapy.

It is planned that up to a total of 12 cycles of therapy will be administered for subjects deriving benefit from this regimen. Continuation of therapy for subjects completing 12 cycles of therapy may be considered on a case-by-case basis after discussion with the Principal Investigator.

#### 4.1.13 Subject Evaluability and Replacement

In the escalation phase, subjects who are not considered fully evaluable per protocol for the primary objective of safety and tolerability per Section 4.3 will be replaced. Subjects who have taken 75% or more of the planned IACS-010759 treatment in cycle 1 will be considered evaluable for MTD. Subjects who have taken less than 75% of planned medication in cycle 1, but who came off study due to a DLT will also be considered evaluable.

#### 4.1.14 Safety Monitoring and Study Stopping Rules

Safety monitoring, including analysis of PK, will be performed by a Safety Monitoring Committee, consisting of the Principal Investigator (and co-investigators as needed) and sponsor representatives (e.g., a designee from the IND Office) and the study-specific Medical Monitor. Additional investigators and staff shall participate in reviews as indicated.

An Independent Data Monitoring Board will not be utilized for this open label study.

#### 4.1.14.1 *Study Stopping Rules*

The Safety Monitoring Committee has the right to recommend to terminate or alter the study design of this clinical study at any time. The principal investigator will be involved in any decisions regarding terminating the study, temporarily suspending enrollment, or stopping ongoing treatment with study treatment. MD Anderson/IND Office (as the sponsor) has the right to terminate the clinical study at any time.

Reasons for terminating the clinical study or a study site's participation include, but are not limited to, the following:

- The incidence or severity of an adverse reaction related to treatment in this study or other studies indicates a potential health hazard to subjects
- Data recording is significantly inaccurate or incomplete
- Study site personnel are noncompliant with study procedures

#### 4.1.14.2 Protocol Violations and Deviations

Protocol violations are defined as significant departures from protocol-required processes or procedures that affect subject safety or benefit potential, or confound assessments of safety or clinical activity. A protocol deviation is a departure from the protocol that does not meet the above criteria. Protocol violations or deviations may be grouped into the following classes:

- Enrollment criteria
- Study activities (missed evaluations or visits) except for those allowed per protocol
- Noncompliance with dose or schedule, including dose calculation, administration, interruption, reduction, or delay; or discontinuation criteria
- Investigational product handling, including storage and accountability
- Informed consent and ethical issues

Every effort will be made to adhere to the schedule of events and all protocol requirements. Variations in schedule of events and other protocol requirements that do not affect the rights and safety of the subject will not be considered as deviations. Such variations may include laboratory assessments completed outside of schedule, occasional missed required research samples such as correlative assays.

#### 4.1.15 Follow-Up at Treatment Discontinuation or Early Withdrawal

Subjects who discontinue treatment for any reason should complete end-of-treatment procedures when possible. End of treatment procedures will include a physical examination, CBC with differential and platelets and chemistry. A bone marrow aspiration may be recommended only if non-response or progressive disease cannot be unequivocally diagnosed from peripheral blood. Although treatment will be discontinued at that time, all subjects who do not die, withdraw consent for follow-up, or become lost to follow-up, will remain on study for

follow-up evaluations. Subject will be followed for possible delayed emergence of IACS-010759 related toxicity at least 30 days after the last protocol treatment. Subjects who discontinue the study will be requested to return for additional PK and/or PD blood daws, approximately every 4 days, when possible, for up to 4 weeks after the last study drug administration to further explore the PK and PD activity of IACS-010759 following discontinuation of study drug. The 30-day (+/-7 days) follow-up visit will be scheduled as a clinic visit for clinical evaluation and physical examinations. If the subject cannot make it to the site for this visit, the required follow up treatment procedures may be performed by a local physician and the records forwarded to the site. The research nurse will also contact the subject by telephone and obtain a verbal assessment of the subject's condition. The phone conversation will then be documented in the subject's charts.

#### 4.1.16 Long-Term Follow-Up

Subjects who achieve any response will be followed for overall survival and response duration for up to 12 cycles. Patients who are responding well to therapy may continue therapy beyond 12 cycles after approval from the PI and sponsor.

If the disease appears to be responding to the study drug, a member of the study staff will call the subject once every 3-6 months for up to 5 years to assess the subject's health.

# 4.2 Study Flowcharts

| Cohorts 1 and 2 | Screen | | | | | | Cycle<br>28 day | | | | | | | Cycl<br>(21 d | | | | cle 3<br>days) | Су | tional<br>cles<br>days) | End of Study<br>or Early<br>Termination |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | -7 to<br>-1 | 1*+ | 2* | 4 | 8* | 9* | 10* | 12* | 14* | 17 | 22 | 28 | 29 | 36 | 42 | 49 | 50 | 70 | Every | 21 days | 30 after<br>last Dose |
| Name of Cycle Day | | C1<br>D1 | C1<br>D2 | C1<br>D4 | C1<br>D8 | C1<br>D9 | C1<br>D10 | C1<br>D12 | C1<br>D14 | C1<br>D17 | C1<br>D22 | C1D<br>28 | C2<br>D1 | C2<br>D8 | C2<br>D14 | C2<br>D21 | C3<br>D1 | C3<br>D21 | CX<br>D20 | CX<br>D21 | 51 |
| +/- days allowable | | | | | | | | | | 1 | 1 | 1 | 2 | 2 | 2 | 2 | 3 | 3 | 4 | 4 | 7 |
| Study Drug§ | | Х | | | Х | Х | Х | Χ | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Disease Assessment | | | | | | | | | | | | | | | | | | | | | |
| Bone marrow aspirate and/or biopsy¥ | Х | | | | | | | | | | | Х | | | | | | х | Every<br>2-3<br>cycle | | х |
| Overall Response Rate <sup>‡</sup> | | | | | | | | | | | | Х | | | | | | Х | , | X <sup>‡</sup> | Х |
| Study Procedures & Examinations | | | | | | | | | | | | | | | | | | | | | |
| Eligibility Assessment & Informed Consent | Х | | | | | | | | | | | | | | | | | | | | |
| Demographics <sup>A</sup> | Х | | | | | | | | | | | | | | | | | | | | |
| Medical history <sup>B</sup> | Х | | | | | | | | | | | | | | | | | | | | |
| MUGA/ECHO | Х | | | | | | | | | | | | | | | | | | | | |
| 12-lead ECG (QTcF) | Х | X <sup>2</sup> | | | Х | | | | X <sup>2</sup> | | Х | X <sup>2</sup> | | | | | | | | | |
| Phys. Exam (inc. weight) | Х | Х | | | Х | | Х | | Х | Χ | Х | Х | Х | | | Х | Х | Х | | Х | Х |
| ECOG | Х | Х | | | | | | | | | | | Х | | | | Х | | | Х | Х |
| Vital Signs (Temp., HR, BP, RR) | Х | X <sup>2</sup> | X <sup>4</sup> | X <sup>5</sup> | X <sup>2</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>2</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>2</sup> | X <sup>3</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>3</sup> | | Х | Х |
| Concomitant Medication <sup>C</sup> | Х | Х | Х | Χ | Х | Χ | Х | Χ | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | | Х | Х |
| Adverse Events <sup>D</sup> | | Х | Х | Х | Х | Х | Х | Χ | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | | Х | Х |
| Labs | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy test | Х | | | | | | | | | | | | | | | | | | | | |
| Blood Hematology <sup>E, I, J</sup> | Х | X <sup>1</sup> | | | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | Χ | Х | Х | Х | | | Х | Х | Х | | Х | Х |
| Chemistry <sup>F, I</sup> | Х | X <sup>1</sup> | | | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | Χ | Х | Х | Х | X <sup>6</sup> | X <sup>6</sup> | Х | Х | Х | | Х | Х |
| Coagulation, lipase, amylase & urinalysis <sup>G, I</sup> | Х | X <sup>1</sup> | | | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | Х | Х | Х | Х | X <sup>6</sup> | X <sup>6</sup> | Χ | | | | Х | Х |
| Lactate and blood pH I, K | Х | X <sup>1</sup> | X <sup>4</sup> | X <sup>5</sup> | X <sup>1</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>3</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>3</sup> | | Х | Х |
| Research Labs | | | | | | | | | | | | | | | | | | | | | |
| Blood collection- pharmacodynamics <sup>H</sup> | Х | X <sup>1</sup> | | | X <sup>1</sup> | | X <sup>1</sup> | | X <sup>1</sup> | | X <sup>1</sup> | X <sup>1</sup> | | | | | | | | | Χ <sup>L</sup> |
| Research Bone marrow aspirate/or biopsy | Х | | | | | | | | | | | Х | | | | | | | | | |

Notes and abbreviations provided on following page.

- + Subjects enrolled in the Food Effect group will consume a high fat meal within 30 minutes prior to study drug administration on Day 1 blood sample collection.
- § Study drug will be administered without food, at least 1 hour before and at least 2 hours after eating, with the exception of Day 1 of Cycle 1 for subjects enrolled in the Food Effect group.
- ¥ Bone marrow aspirate/biopsy will be performed as clinically indicated, at least once every 3 cycles.
- ‡ Overall Response Rate (ORR) assessment will be performed on the same schedule as bone marrow aspirate/biopsy (every 2-3 cycles during additional cycles). ORR definitions are provided in Section 5.2.2.

<sup>&</sup>lt;sup>A</sup> including Date of Birth; sex; height; race; ethnicity

<sup>&</sup>lt;sup>B</sup> including oncology history, radiation history

<sup>&</sup>lt;sup>c</sup> name, indication, dose, route, start and end dates

<sup>&</sup>lt;sup>D</sup> starting or worsening after study drug administration (signs and symptoms occurring prior to the first dose of study medication on Day 1 should be recorded under the subject's Medical History).

<sup>&</sup>lt;sup>E</sup> complete blood count, differential, platelets

<sup>&</sup>lt;sup>F</sup> glucose, total protein, albumin, electrolytes [sodium, potassium, chloride, total CO₂], calcium, phosphorus, magnesium, uric acid, bilirubin (total, direct), SGPT (ALT) or SGOT (AST), alkaline phosphatase, creatinine, blood urea nitrogen, CPK

<sup>&</sup>lt;sup>G</sup> PT, PTT, fibrinogen, INR

<sup>&</sup>lt;sup>H</sup>Oxygen consumption, metabolites, protein, mRNA analysis

<sup>&</sup>lt;sup>1</sup> To be performed weekly during the first cycle of the increased dose for any intra-subject dose escalation

<sup>&</sup>lt;sup>1</sup> For purposes of data collection, test results below the limit of quantitation will be reported as "0"

<sup>&</sup>lt;sup>k</sup> If the Investigator determines that the dose of study drug should be interrupted, additional PK, lactate and blood pH assessments will be collected pre-dose (within 2 hours of dosing) and 6 hours +/- 30 minutes post study drug administration upon resumption of dosing. If the dose of study drug is reduced, additional PK assessments will be collected pre-dose (within 2 hours of dosing) and 2, 4, 6, 8, 12 (+/- 15 mins) and 72 hours (+/- 4 hours) after starting the reduced study drug dose.

<sup>&</sup>lt;sup>L</sup> Additional PK and/or PD draws from peripheral blood may be obtained ~every 4 days, when possible, for up to 4 weeks after last study drug administration in subjects who discontinue the study.

<sup>&</sup>lt;sup>M</sup> In addition to the time points indicated in the Table, additional draws from peripheral blood for PK analysis may be obtained during Cycle 2 and beyond at the discretion of the Investigator.

<sup>&</sup>lt;sup>1</sup> collected pre-dose (within 2 hours of dosing) and 6 hours +/- 30 minutes post study drug administration

<sup>&</sup>lt;sup>2</sup> collected pre-dose (within 2 hours of dosing) and 2, 4, 6, 8 and 12 hours (+/- 15 mins) post study drug administration

<sup>&</sup>lt;sup>3</sup> collected pre-dose (within 2 hours of dosing)

<sup>&</sup>lt;sup>4</sup> collected 24 hours +/- 2 hours post study drug administration

<sup>&</sup>lt;sup>5</sup> collected 72 hours +/- 4 hours post study drug administration

<sup>&</sup>lt;sup>6</sup> collected pre-dose

<sup>\*</sup> Treatment will be administered as an inpatient for 24 hours on Day 1 of Cycle 1 and then starting again on Day 8 for the next 7 days.

## Cohorts 3-4 Dose-Escalation

| Conorts 5-4 Dose-Escalation | Screen | | | | | Cycle<br>21 da | | | | | | | Cycle 2<br>21 day: | | | Сус<br>(21 с | | Addition<br>Cyclo<br>(21 da | es | End of Study<br>or Early<br>Termination |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | -7 to<br>-1 | 1+ | 2 | 4 | 7* | 8 | 12 | 15 | 17 | 21 | 22 | 29 | 36 | 37 | 42 | 43 | 63 | Every 2 | 1 days | 30 after<br>last Dose |
| Name of Cycle Day | | C1<br>D1 | C1<br>D2 | C1<br>D4 | C1<br>D7 | C1<br>D8 | C1<br>D12 | C1<br>D15 | C1<br>D17 | C1<br>D21 | C2<br>D1 | C2<br>D8 | C2<br>D15 | C2<br>D16 | C2<br>D21 | C3<br>D1 | C3<br>D21 | CX<br>D20 | CX<br>D21 | 51 |
| +/- days allowable | | | | 1 | 1 | 1 | 1 | 1 | 2 | +2 | 1 | 1 | 1 | 2 | 1 | 3 | 3 | 4 | 4 | 7 |
| Study Drug§ | | I | NDU | CTIOI | V | | | | | | | | М | AINTE | NANC | E | | | | |
| Study Drugg | | Х | Х | Х | Х | Х | | Х | | | Х | Х | Х | | | Х | | | | |
| Disease Assessment | | | | | | | | | | | | | | | | | | | | |
| Bone marrow aspirate and/or biopsy¥ | х | | | | | | | | | х | | | | | | | Х | Every 2-3<br>cycle | | x |
| Overall Response Rate <sup>‡</sup> | | | | | | | | | | Х | | | | | | | Х | | Χ‡ | Х |
| Study Procedures & Examinations | | | | | | | | | | | | | | | | | | | | |
| Eligibility Assessment & Informed Consent | Х | | | | | | | | | | | | | | | | | | | |
| Demographics <sup>A</sup> | Х | | | | | | | | | | | | | | | | | | | |
| Medical history <sup>B</sup> | Х | | | | | | | | | | | | | | | | | | | |
| MUGA/ECHO | Х | | | | | | | | | | | | | | | | | | | |
| Dilated eye exam with fundus photos <sup>N</sup> | | Х | | | | | | | | | | | | | | | | | | |
| Neurology review and exam <sup>0</sup> | | Х | | | | | | | | | | | | | | | | | | |
| 12-lead ECG (QTcF) | Х | X <sup>2</sup> | | | X <sup>1</sup> | | | X <sup>1</sup> | | Х | | | | | | | | | | |
| Phys. Exam (inc. weight) | Х | Х | | | Х | | | Х | | Х | Х | | | | Х | Х | Х | | Х | Х |
| ECOG | Х | Х | | | | | | | | | Х | | | | | Х | | | Х | Х |
| Vital Signs (Temp., HR, BP, RR) | Х | X <sup>2</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>2</sup> | X <sup>1</sup> | Х | X <sup>1</sup> | | Χ | X <sup>3</sup> | X <sup>3</sup> | X <sup>1</sup> | Х | Х | X <sup>3</sup> | Х | | Х | X |
| Concomitant Medication <sup>C</sup> | Х | Х | Χ | Х | Х | Х | Χ | Х | Х | Χ | Х | Х | Χ | Х | Х | Х | Х | | Χ | X |
| Adverse Events <sup>D</sup> | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | | Х | X |
| Labs | | | | | | | | | | | | | | | | | | | | |
| Pregnancy test | X | | | | | | | | | | | | | | | | | | | |
| Blood Hematology <sup>E, I, J</sup> | Х | X <sup>1</sup> | | | X <sup>3</sup> | X <sup>3</sup> | Х | X <sup>3</sup> | Х | Х | Х | | | Х | Х | Х | Х | | Х | X |
| Chemistry <sup>F, I</sup> | Х | X <sup>1</sup> | | | X <sup>3</sup> | X <sup>3</sup> | Х | X <sup>3</sup> | Х | Х | Х | X <sup>3</sup> | X <sup>3</sup> | Х | Х | Х | Х | | Х | X |
| Coagulation, lipase, amylase & urinalysis G, I | Х | X <sup>1</sup> | | | X <sup>3</sup> | X <sup>3</sup> | Х | X <sup>3</sup> | Х | Х | Х | X <sup>3</sup> | X <sup>3</sup> | Х | Х | | | | Х | Х |
| Lactate and blood pH I, K | Х | X <sup>1</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>1</sup> | X <sup>1</sup> | Х | X <sup>1</sup> | Χ | Х | X <sup>3</sup> | X <sup>3</sup> | X <sup>1</sup> | Х | Х | X <sup>3</sup> | Х | | Х | Х |
| Research Labs | | | | | | | | | | | | | | | | | | | | |

| Blood collection- pharmacodynamics <sup>H</sup> | X | X <sup>1</sup> | | | X <sup>1</sup> | | | X <sup>1</sup> | | Χ | | | | | | | | | $X^L$ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Research Bone marrow aspirate/or biopsy | Х | | | | | | | | | Χ | | | | | | | | | |
| Pharmacokinetics Blood samples I,K,M | | X <sup>2</sup> | <b>X</b> <sup>3</sup> | X <sup>3</sup> | X <sup>2</sup> | X <sup>1</sup> | Х | X <sup>1</sup> | Х | Х | X <sup>3</sup> | X <sup>3</sup> | X <sup>2</sup> | Х | Х | X <sup>3</sup> | Х | Х | X <sup>L</sup> |

Notes and abbreviations provided on following page.

<sup>&</sup>lt;sup>A</sup> including Date of Birth; sex; height; race; ethnicity

<sup>&</sup>lt;sup>B</sup> including oncology history, radiation history

<sup>&</sup>lt;sup>c</sup> name, indication, dose, route, start and end dates

<sup>&</sup>lt;sup>D</sup> starting or worsening after study drug administration (signs and symptoms occurring prior to the first dose of study medication on Day 1 should be recorded under the subject's Medical History).

<sup>&</sup>lt;sup>E</sup> complete blood count, differential, platelets

<sup>&</sup>lt;sup>F</sup> glucose, total protein, albumin, electrolytes [sodium, potassium, chloride, total CO₂], calcium, phosphorus, magnesium, uric acid, bilirubin (total, direct), SGPT (ALT) or SGOT (AST), alkaline phosphatase, creatinine, blood urea nitrogen, CPK

<sup>&</sup>lt;sup>G</sup> PT, PTT, fibrinogen, INR

<sup>&</sup>lt;sup>H</sup>Oxygen consumption, metabolites, protein, mRNA analysis

<sup>&</sup>lt;sup>1</sup> To be performed weekly during the first cycle of the increased dose for any intra-subject dose escalation

<sup>&</sup>lt;sup>1</sup> For purposes of data collection, test results below the limit of quantitation will be reported as "0"

<sup>&</sup>lt;sup>K</sup> If the Investigator determines that the dose of study drug should be interrupted, additional PK, lactate and blood pH assessments will be collected pre-dose (within 2 hours of dosing) and 4 hours +/- 30 minutes post study drug administration upon resumption of dosing; additional PK assessments may be performed during the interruption at the description of the Investigator. If the dose of study drug is reduced, additional PK assessments will be collected pre-dose (within 2 hours of dosing) prior to starting the reduced study drug dose. Additional unscheduled PK, lactate and pH blood draws may be collected per PI judgement when indicated for further safety follow-up.

<sup>&</sup>lt;sup>L</sup>Additional PK and/or PD draws from peripheral blood may be obtained ~every 4 days, when possible, for up to 4 weeks after last study drug administration in subjects who discontinue the study.

<sup>&</sup>lt;sup>M</sup> In addition to the time points indicated in the Table, additional draws from peripheral blood for PK analysis may be obtained at the discretion of the Investigator.

<sup>&</sup>lt;sup>N</sup> Baseline dilated eye exam with fundus photos, including distance acuity (visual acuity charts using refraction-based visual acuity measurement), ophthalmoscopy and slit lamp exam, may be performed up to 14 days prior to study drug administration.

<sup>&</sup>lt;sup>o</sup> Baseline neurology review and exam to be performed by consultant neurologist up to 14 days prior to study drug administration. The baseline neurology exam may include, but is not limited to, gait and station, cerebellar functions (coordination), upper and lower extremity reflexes, upper and lower muscle strength and sensation.

<sup>&</sup>lt;sup>1</sup> collected pre-dose (same calendar day of dosing) and 4 hours +/- 30 minutes post study drug administration

<sup>&</sup>lt;sup>2</sup> collected pre-dose (same calendar day of dosing) and 2, 4, 6, 8 hours (+/- 30 mins) post study drug administration. Note: vitals may be collected (+/- 60 mins) post study drug administration.

<sup>&</sup>lt;sup>3</sup> collected pre-dose (same calendar day of dosing)

- \* Treatment will be administered as an inpatient for 24 hours on Day 7 of Cycle 1.
- + Subjects enrolled in the Food Effect group will consume a high fat meal within 30 minutes prior to study drug administration on Day 1 blood sample collection. § Study drug will be administered without food, at least 1 hour before and at least 2 hours after eating, with the exception of Day 1 of Cycle 1 for subjects enrolled in the Food Effect group. Induction or maintenance doses and alternative duration of induction doses or other maintenance schedules of IACS-010759, not to exceed 6 mg, may be pursued depending on the safety and PK/PD data observed.
- ¥ Bone marrow aspirate/biopsy will be performed as clinically indicated, at least once every 3 cycles.
- ‡ Overall Response Rate (ORR) assessment will be performed on the same schedule as bone marrow aspirate/biopsy (every 2-3 cycles during additional cycles). ORR definitions are provided in Section 5.2.2.


Cohorts 5-6 Dose-Escalation and Cohort 7 Dose-Expansion

| | Screen | | | | | Cycle<br>21 da | | | | | | | Cycle 2<br>21 day: | | | Cyc<br>(21 d | | Additio<br>Cycle<br>(21 da | es | End of Study<br>or Early<br>Termination |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | -7 to<br>-1 | 1+ | 2 | 4 | 5* | 8 | 12 | 15 | 17 | 21 | 22 | 29 | 36 | 37 | 42 | 43 | 63 | Every 2 | L days | 30 after<br>last Dose |
| Name of Cycle Day | | C1<br>D1 | C1<br>D2 | C1<br>D4 | C1<br>D5 | C1<br>D8 | C1<br>D12 | C1<br>D15 | C1<br>D17 | C1<br>D21 | C2<br>D1 | C2<br>D8 | C2<br>D15 | C2<br>D16 | C2<br>D21 | C3<br>D1 | C3<br>D21 | CX<br>D20 | CX<br>D21 | 51 |
| +/- days allowable | | | | 1 | | | 1 | 1 | 2 | +2 | 1 | 1 | 1 | 2 | 1 | 3 | 3 | 4 | 4 | 7 |
| Study Drug§ | | II | NDUC | CTION | <b>J</b> P | | | | | | | MA | INTEN | ANCE <sup>P</sup> | | | | | | |
| Disease Assessment | | | | | | | | | | | | | | | | | | | | |
| Bone marrow aspirate and/or biopsy¥ | Х | | | | | | | | | Х | | | | | | | х | Every 2-3<br>cycle | | Х |
| Overall Response Rate <sup>‡</sup> | | | | | | | | | | Х | | | | | | | Х | | X <sup>‡</sup> | Х |
| Study Procedures & Examinations | | | | | | | | | | | | | | | | | | | | |
| Eligibility Assessment & Informed Consent | Х | | | | | | | | | | | | | | | | | | | |
| Demographics <sup>A</sup> | Х | | | | | | | | | | | | | | | | | | | |
| Medical history <sup>B</sup> | Х | | | | | | | | | | | | | | | | | | | |
| MUGA/ECHO | Х | | | | | | | | | | | | | | | | | | | |
| Dilated eye exam with fundus photos <sup>N</sup> | | Х | | | | | | | | | | | | | | | | | | |
| Neurology review and exam <sup>o</sup> | | Х | | | | | | | | | | | | | | | | | | |
| 12-lead ECG (QTcF) | Х | X <sup>2</sup> | | | X <sup>1</sup> | | | X <sup>1</sup> | | Х | | | | | | | | | | |
| Phys. Exam (inc. weight) | Х | Х | | | Х | | | Х | | Х | Х | | | | Х | Х | Х | | Х | Х |
| ECOG | Х | Х | | | | | | | | | Х | | | | | Х | | | Х | Х |
| Vital Signs (Temp., HR, BP, RR) | Х | X <sup>2</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>2</sup> | X <sup>1</sup> | Х | X <sup>1</sup> | | Х | X <sup>3</sup> | X <sup>3</sup> | X <sup>1</sup> | Х | Х | X <sup>3</sup> | Х | | Х | Х |
| Concomitant Medication <sup>C</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | Х | Х |
| Adverse Events <sup>D</sup> | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | Х | Х |
| Labs | | | | | | | | | | | | | | | | | | | | |
| Pregnancy test | Х | | | | | | | | | | | | | | | | | | | |
| Blood Hematology <sup>E, I, J</sup> | Х | X <sup>1</sup> | | | X <sup>3</sup> | X <sup>3</sup> | Х | X <sup>3</sup> | Χ | Х | Х | | | Х | Х | Х | Х | | Х | Х |
| Chemistry <sup>F, I</sup> | Х | X <sup>1</sup> | | | X <sup>3</sup> | X <sup>3</sup> | Х | X <sup>3</sup> | Χ | Х | Х | X <sup>3</sup> | X <sup>3</sup> | Х | Х | Х | Х | | Х | Х |
| Coagulation, lipase, amylase & urinalysis <sup>G, I</sup> | Х | X <sup>1</sup> | | | X <sup>3</sup> | X <sup>3</sup> | Х | X <sup>3</sup> | Х | Х | Х | X <sup>3</sup> | X <sup>3</sup> | Х | Х | | | | Х | Х |
| Lactate and blood pH I, K | Х | X <sup>1</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>1</sup> | X <sup>1</sup> | Х | X <sup>1</sup> | Χ | Х | X <sup>3</sup> | X <sup>3</sup> | X <sup>1</sup> | Х | Х | X <sup>3</sup> | Х | | Х | Х |
| Research Labs | | | | | | | | | | | | | | | | | | | | |
| Blood collection- pharmacodynamics <sup>H</sup> | Х | X <sup>1</sup> | | | X <sup>1</sup> | | | X <sup>1</sup> | | Х | | | | | | | | | | Χ <sup>L</sup> |

| Research Bone marrow aspirate/or biopsy | X | | | | | | | | | Х | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Pharmacokinetics Blood samples I,K,M | | X <sup>2</sup> | X <sup>3</sup> | X <sup>3</sup> | X <sup>4</sup> | X <sup>1</sup> | Χ | X <sup>1</sup> | Χ | Χ | $X_3$ | X <sup>3</sup> | X <sup>2</sup> | Χ | Χ | X <sup>3</sup> | Χ | Х | $X^{L}$ |

Notes and Abbreviations:

<sup>&</sup>lt;sup>A</sup> including Date of Birth; sex; height; race; ethnicity

<sup>&</sup>lt;sup>B</sup> including oncology history, radiation history

<sup>&</sup>lt;sup>c</sup> name, indication, dose, route, start and end dates

<sup>&</sup>lt;sup>D</sup> starting or worsening after study drug administration (signs and symptoms occurring prior to the first dose of study medication on Day 1 should be recorded under the subject's Medical History).

<sup>&</sup>lt;sup>E</sup> complete blood count, differential, platelets

<sup>&</sup>lt;sup>F</sup> glucose, total protein, albumin, electrolytes [sodium, potassium, chloride, total CO₂], calcium, phosphorus, magnesium, uric acid, bilirubin (total, direct), SGPT (ALT) or SGOT (AST), alkaline phosphatase, creatinine, blood urea nitrogen, CPK

<sup>&</sup>lt;sup>G</sup> PT, PTT, fibrinogen, INR

<sup>&</sup>lt;sup>H</sup>Oxygen consumption, metabolites, protein, mRNA analysis

<sup>&</sup>lt;sup>1</sup> To be performed weekly during the first cycle of the increased dose for any intra-subject dose escalation

<sup>&</sup>lt;sup>1</sup> For purposes of data collection, test results below the limit of quantitation will be reported as "0"

<sup>&</sup>lt;sup>K</sup> If the Investigator determines that the dose of study drug should be interrupted, additional PK, lactate and blood pH assessments will be collected pre-dose (within 2 hours of dosing) and 4 hours +/- 30 minutes post study drug administration upon resumption of dosing; additional PK assessments may be performed during the interruption at the description of the Investigator. If the dose of study drug is reduced, additional PK assessments will be collected pre-dose (within 2 hours of dosing) prior to starting the reduced study drug dose. Additional unscheduled PK, lactate and pH blood draws may be collected per PI judgement when indicated for further safety follow-up.

<sup>&</sup>lt;sup>L</sup> Additional PK and/or PD draws from peripheral blood may be obtained ~every 4 days, when possible, for up to 4 weeks after last study drug administration in subjects who discontinue the study.

<sup>&</sup>lt;sup>M</sup> In addition to the time points indicated in the Table, additional draws from peripheral blood for PK analysis may be obtained at the discretion of the Investigator.

<sup>&</sup>lt;sup>N</sup> Baseline dilated eye exam with fundus photos, including distance acuity (visual acuity charts using refraction-based visual acuity measurement), ophthalmoscopy and slit lamp exam, may be performed up to 14 days prior to study drug administration.

<sup>&</sup>lt;sup>o</sup> Baseline neurology review and exam to be performed by consultant neurologist up to 14 days prior to study drug administration. The baseline neurology exam may include, but is not limited to, gait and station, cerebellar functions (coordination), upper and lower extremity reflexes, upper and lower muscle strength and sensation.

<sup>&</sup>lt;sup>P</sup> The dose regimen for the induction and maintenance doses are provided in Table 2.

<sup>&</sup>lt;sup>1</sup> collected pre-dose (same calendar day of dosing) and 4 hours +/- 30 minutes post study drug administration

<sup>&</sup>lt;sup>2</sup> collected pre-dose (same calendar day of dosing) and 2, 4, 6, 8 hours (+/- 30 mins) post study drug administration. Note: vitals may be collected (+/- 60 mins) post study drug administration.

<sup>&</sup>lt;sup>3</sup> collected pre-dose (same calendar day of dosing)

<sup>&</sup>lt;sup>4</sup> collected pre-dose (same calendar day of dosing) and 2, 4, 6, 8 hours (+/- 30 mins) and 24 hours (+/- 2 hours) post study drug administration. Note: vitals may be collected (+/- 60 mins) post study drug administration.
- \* Treatment will be administered as an inpatient for 24 hours on Day 5 of Cycle 1.
- + Subjects enrolled in the Food Effect group will consume a high fat meal within 30 minutes prior to study drug administration on Day 1 blood sample collection. § Study drug will be administered without food, at least 1 hour before and at least 2 hours after eating, with the exception of Day 1 of Cycle 1 for subjects enrolled in the Food Effect group. Induction or maintenance doses and alternative duration of induction doses or other maintenance schedules of IACS-010759, not to exceed 6 mg, may be pursued depending on the safety and PK/PD data observed.
- ¥ Bone marrow aspirate/biopsy will be performed as clinically indicated, at least once every 3 cycles.
- ‡ Overall Response Rate (ORR) assessment will be performed on the same schedule as bone marrow aspirate/biopsy (every 2-3 cycles during additional cycles). ORR definitions are provided in Section 5.2.2.

IACS2015-001: Protocol Amendment #11 (01-21-20) 

### Study Objectives & Endpoints

| Primary Objectives | Safety & Tolerability |
|---|---|
| | Determine Dose Limiting Toxicities |
| | Establish MTD and RP2D |
| <b>Secondary Objectives</b> | IACS-010759 pharmacokinetics and food effect |
| | Preliminary Clinical Efficacy (overall response rates, duration of |
| | response, progression-free survival, overall survival) |
| <b>Exploratory objectives</b> | Pharmacodynamic and exploratory biomarkers of activity of IACS- |
| | 010759 |

Clinical study data will be entered into Medidata Rave, the clinical data base, via electronic case report forms. The Statistical Analysis Plan (SAP) will include detailed and specific description of all analysis to be performed on the clinical data from this study. The SAP will be finalized prior to database lock.

All statistical analyses will be performed using Version 9.4 or later of Statistical Analysis Software (SAS®). Data summaries will use descriptive statistics (number of subjects [n], mean, standard deviation [SD], Q1, median, Q3, minimum, and maximum) for continuous variables, and frequency and percentage for categorical and ordinal variables. If there are missing values, the number missing will be presented, but without a percentage. All data collected will be included in by-subject data listings.

Unless otherwise specified, all tests will be two-tailed using a 0.05 level of significance. All confidence intervals (CIs) will be two-sided 95% confidence intervals.

All subjects who received any study drug and who had any on-treatment evaluation will be included in the Full Analysis Set (FAS).

### 4.3 Safety and tolerability

### 4.3.1 Endpoints & Assessment Methods

Laboratory tests, vital sign measurements, physical exams and subject interviews will be performed to detect new abnormalities and deteriorations of any pre-existing conditions. All "treatment-emergent" clinically significant abnormalities and deteriorations that begin or worsen in severity after initial administration of IACS-010759 and documented as such in the medical records should be recorded in the Case Report Forms as Adverse Events and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.03.

The MTD will be determined in accordance with Section 4.1.7.

### 4.3.2 Subject Evaluation & Statistics

The FAS will be used for evaluation of safety.

Adverse events will be coded using the MedDRA dictionary. Incidences of treatment-emergent adverse events (TEAE, those events that started after dosing or worsened in severity after dosing) will be presented overall and by maximum severity (according to CTCAE Ver 4.03) and relationship to study medication.

For each continuous laboratory parameter, results will be categorized as low, normal, or high based on the laboratory normal ranges. Frequencies and percentages will be presented by cohort for the shifts in these categories (i.e., low to normal, low to high, high to low, etc.) from baseline to each post-treatment assessment time point. Additionally, for each continuous hematology and chemistry parameter, descriptive statistics will be presented by cohort for the changes from baseline to each post-treatment assessment time point. Descriptive statistics will be presented by cohort for the changes in vital signs from baseline to each post-treatment assessment time point.

### 4.4 Clinical Efficacy

### 4.4.1 Subject Evaluation & Statistics

The FAS will be the basis for the evaluation of clinical efficacy.

Disease assessment will be performed at the end of Cycles 1, 3, and thereafter every 2-3 cycles at the discretion of the treating physician. While the bone marrow aspirate/biopsy will be performed as clinically indicated, testing will occur at least once every 3 cycles.

Descriptive statistics will be provided for continuous variables and frequency tables will be used to summarize categorical variables. The Overall Response Rate and the proportions of subjects who experienced CR, Cri, PR, MLFS (morphologic leukemia-free state), hematologic improvements, Recurrence of Disease (RD) and Best Response measurement along with the corresponding exact 95% confidence intervals will be displayed.

Kaplan-Meier method will be used to estimate the duration of response, progression-free survival and overall survival. These time to event variables will be summarized using the 25<sup>th</sup> percentile, Median, and 75<sup>th</sup> percentile as well as the minimum and maximum time to event, calculated by Kaplan-Meier method, and will be displayed graphically.

#### 4.4.2 Endpoints & Assessment Methods

Objective Overall Response Rate (ORR) for subjects with AML include CR, CRi, PR and morphologic leukemia-free state [22] with or without cytogenetic response and hematologic improvements. The responses are defined as below:

### Complete Remission (CR)

For subjects to be classified as being in CR, they must have bone marrow regenerating normal hematopoietic cells and achieve a morphologic leukemia-free state and must have an ANC >  $1 \times 10^9$ /L and platelet count  $\ge 100 \times 10^9$ /L, and normal marrow differential with < 5% blasts, and subjects will be red blood cell (RBC) and platelet transfusion independent (defined as 4 weeks without RBC transfusion and 1 week without platelet transfusion). There should be no evidence of extramedullary leukemia.

Complete Remission with Incomplete Hematological Recovery (CRi)
 For subjects to be classified as being in CRi, they must fulfill the criteria for CR except for incomplete hematological recovery with residual neutropenia (ANC ≤ 1 × 10<sup>9</sup>/L) with or without thrombocytopenia (platelet count < 100 × 10<sup>9</sup>/L). In addition, subjects do not need to be RBC or platelet transfusion independent (modification to Cheson criteria).

#### • Partial Remission (PR)

For subjects to be classified as being in PR, they must have bone marrow regenerating normal hematopoietic cells with evidence of peripheral recovery with no (or only a few

regenerating) circulating blasts and with a decrease of at least 50% in the percentage of blasts in the bone marrow aspirate with the total marrow blasts between 5% and 25%.

### • Morphologic leukemia-free state (MLFS):

Bone marrow: ≤5% myeloblasts

#### Hematologic Improvement (HI):

Hematologic response must be described by the number of positively affected cell lines.

- Erythroid response (E) (pretreatment Hgb <11 g/dL)</li>
- Hgb increase by ≥1.5 g/dL
- Platelet response (P) (pretreatment platelets <100 x10<sup>9</sup>/L)
- Absolute increase of  $\ge 30 \times 10^9$ /L for subjects starting with  $> 20 \times 10^9$ /L platelets
- $\circ$  Increase from < 20 x 10<sup>9</sup>/L to > 20 x 10<sup>9</sup>/L and by at least 100%
- Neutrophil response (N) (pretreatment ANC <1.0 x10<sup>9</sup>/L)
- o At least 100% increase and an absolute increase > 0.5 x 10<sup>9</sup>/L
- Blast response (B)≥50% reduction in peripheral blood or bone marrow blasts but still >5%

### • Recurrence of Disease (RD)

Relapse after CR is defined as a reappearance of leukemic blasts in the peripheral blood or  $\geq 5\%$  blasts in the bone marrow aspirate not attributable to any other cause or reappearance or new appearance of extramedullary leukemia. Relapse after PR is similarly defined with reappearance of significant numbers of peripheral blasts and an increase in the percentage of blasts in the bone marrow aspirate to > 25% not attributable to any other cause or reappearance or new appearance of extramedullary leukemia.

Best Response measurement: Response will be measured and defined for primary endpoints as the best response achieved during the first 3 cycles of therapy, or at time off study, for those subjects discontinuing treatment before the completion of 3 cycles of therapy. Best response is defined to be the best-measured response (ORR=CR+CRp+PR+MLFS) post-treatment up to that time. Best response will also be evaluated for the full treatment period using all assessments up to and including treatment discontinuation.

**Duration of Response**: length of time from the first objective evidence of response to the first objective evidence of disease progression.

**Progression-Free Survival**: length of time (up to 5 years) from the date of first treatment to the first objective evidence of disease progression or death, whichever is earlier.

**Overall Survival**: length of time from the date of first administration of study drug to the date of death from any cause.

### 4.5 IACS-010759 Plasma Drug Levels

#### 4.5.1 Subject Evaluation & Statistics

Only subjects who received at least one dose of IACS-010759, and provided both the baseline sample and at least one post-treatment sample, will be evaluated.

### 4.5.2 Endpoints & Assessment Methods

Collection of samples to assess the plasma concentration of IACS-010759 will be required for all subjects. Peripheral blood (5 mL) will be collected at the time points indicated in section 4.2.

A validated LC-MS/MS bioanalytical method will be used at the MDACC, Institute for Applied Cancer Science (IACS) research labs, located at 4SCRB2.1175, 1901 East Road, Houston, TX to quantify IACS-010759 in human plasma.

Pharmacokinetic parameters will be calculated using Phoenix WinNonlin 6.3 software package.

### 4.6 Biological activity of IACS-010759

### 4.6.1 Subject Evaluation & Statistics

Only subjects who received at least one dose of IACS-010759, and provided the baseline and at least one post-treatment sample, will be evaluated.

PD data will be summarized graphically and with descriptive statistics by time and dose.

### 4.6.2 Endpoints & Assessment Methods

To evaluate PD biomarkers, approximately 30 cc of peripheral blood will be collected in green top tubes and 5 cc of bone marrow will be collected at the time points indicated in section 4.2. Upon isolation of blasts cells, baseline and post-treatment biological activity will be assessed using assays that are informed by preclinical studies using AML cell line and subject derived models. These include but are not limited to:

- Pre and post-treatment measurement of OXPHOS inhibition, using Seahorse Seahorse
   XF bioanalyzer to measure oxygen consumption in blast cells isolated from the peripheral blood.
- Pre and post-treatment measurement of metabolites related to mitochondria metabolism, glycolysis, amino acid and nucleotide biosynthesis, to measure changes that have been associated with inhibition of OXPHOS and response in preclinical models.
- Pre and post treatment measurement of mRNAs using gene expression profiling or other quantitative methods to assess mRNA signatures that has been identified utilizing preclinical models treated with IACS-010759.

Any leftover sample or tissue including bone marrow, if available, will be stored for potential future exploratory research into factors that may influence development of AML and/or response to IACS-010759 (where response is defined broadly to include efficacy, tolerability or safety) or additional exploratory pharmacogenetic evaluations, including RNA microarray analyses or DNA, and xenografting into immunodeficient mice. Excess samples will be stored at MD Anderson Cancer Center, IACS laboratory, located at 4SCR6.1100, 1901 East Road, Houston, TX.

# 5 Subject Eligibility

#### 5.1 Inclusion Criteria

Eligible subjects **must fulfill** all of the following criteria:

1. Subjects with AML should have failed any prior induction therapy regimen or have relapsed after prior therapy (defined as patients in first relapse and less than 12 months from diagnosis [short first remission] or in second or later relapse

Dose-escalation phase: Subjects with confirmed relapsed or refractory AML and no available treatment options with known benefit

Expansion phase: Subjects with relapsed/refractory AML who have failed therapy with up to one prior salvage regimen and no available treatment options with known benefit Exception: stem cell transplant [SCT] or stem cell therapy for subjects who previously underwent SCT/stem cell therapy, and are currently in remission will not be considered a salvage regimen.

- 2. Eastern Cooperative Oncology Group (ECOG) ≤ 2 (see appendix 9.3)
- 3. Patients who have had prior SCT are eligible if they have a relapse > 3 months since autologous or allogeneic stem cell transplantation provided,
  - No clinically significant active graft-versus-host disease (GVHD > grade 1).
  - No treatment with high dose steroids for GVHD (i.e. >20 mg Prednisolone or equivalent per day).
  - No treatment with immunosuppressive drugs with the exception of cyclosporine and tacrolimus.
- 4. Subjects with history of CNS disease are allowed if at the time of day 1 of the study there is no evidence of active CNS disease as documented by negative imaging or spinal fluid analysis carried out at least 2 weeks prior to the first study drug administration in a subject with no clinical signs of CNS disease.
- 5. Adequate renal and hepatic function:
  - Serum creatinine ≤ 2.0 X ULN
  - Total bilirubin  $\leq$  2 times the upper limit of normal (ULN) (or </=3.0 x ULN if deemed to be elevated due to Gilbert's disease or leukemia)
  - ALT and AST ≤ 2.5 times ULN (≤ 5.0 x ULN if due to leukemic involvement).
- 6. Negative urine pregnancy test within 72 hours prior to the first dose of study therapy for women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally post-menopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months).
- 7. Have been informed of other treatment options and is not a candidate for standard treatment options or stem cell transplant at the time of enrollment.
- 8. Age  $\geq$ 18 years.
- 9. In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of IACS-010759 administration will be at least 2 weeks or 5 half-lives (whichever is shorter) for cytotoxic/noncytotoxic agents and biological/immune-based therapies, including investigational agents. The half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochures, or drug-administration manuals) and will be documented in the protocol eligibility document. The use of chemotherapeutic or anti-leukemic agents is not permitted during the study with the following exceptions: (1) intrathecal (IT) therapy for subjects with controlled CNS leukemia at the discretion of the PI and with the agreement of the Sponsor. (2) Use of hydroxyurea for subjects with rapidly proliferative disease is allowed before the start of study therapy and for the first 2 cycles on therapy. These medications will be recorded in the case-report form.

10. Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment.

Adequate methods of contraception include:

- Total abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
- Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
- Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
- Combination of any of the two following (a+b or a+c or b+c)
- Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
- b. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
- c. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository In case of use of oral contraception, women should have been stable on the same pill before taking study treatment.

**Note:** Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction. Women are considered postmenopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

11. Able and willing to give valid written informed consent.

# **5.2 Exclusion Criteria**

Subjects <u>may not</u> enter the study if they fulfill any of the following criteria:

| 1 | Drive exposure to IACS 0107E0 or other exidetive phosphogration labilities |
|---|---|
| 1. | Prior exposure to IACS-010759 or other oxidative phosphorylation Inhibitors. |
| 2. | <ul> <li>Unstable cardiovascular function:</li> <li>Symptomatic ischemia, or</li> <li>Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on antiarrhythmic agents are excluded; 1<sup>st</sup> degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) will not be excluded), or</li> <li>Congestive heart failure (CHF) NYHA Class ≥ 3 (Appendix 9.5), or</li> <li>Myocardial infarction (MI) within 6 months.</li> <li>Left ventricular ejection fraction &lt; 40 %.</li> <li>Hypertension &gt; 160 mm Hg systolic or &gt; 100 mm Hg diastolic with or without antihypertensive therapy.</li> </ul> |
| 3. | Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery from the surgical procedure |
| 4. | Presence of $\geq$ CTCAE grade 2 toxicity (except alopecia or peripheral neuropathy) due to prior cancer therapy. |
| 5. | Known positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV). |
| 6. | Active uncontrolled infection. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines is acceptable. |
| 7. | Participation in any other clinical trial involving another investigational agent for the treatment of AML within 2 weeks prior to day 1 of the study or at least 5 half-lives of the investigational agent, whichever is shorter. |
| 8. | Lactate levels > 2 mmol/L and or and serum pH <7.35 at screening. |
| 9. | Subject currently being treated with biguanides or other agents known to increase risk of lactic acidosis (reference Appendix 10.1). |
| 10. | Subject has significant gastrointestinal abnormalities, including ulcerative colitis, chronic diarrhea associated with intestinal malabsorption, Crohn's disease, and/or prior surgical procedures affecting absorption or requirement for intravenous (IV) alimentation. |
| 11. | Subjects with uncontrolled Type I or II diabetes mellitus |
| 12. | Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study. |
| 13. | Women who are breast-feeding or pregnant as evidenced by positive urine pregnancy test done within 72 hours of first dosing. |
| 14. | Subject has a concurrent active malignancy under treatment, with the exception of: -Adequately treated carcinoma in situ of the breast or cervix uteri -Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin -Low-grade, early-stage prostate cancer with no requirement for therapy -Previous malignancy confined |
| 15. | Acute promyelocytic leukemia. |

IACS2015-001: Protocol Amendment #11 (01-21-20)

- 16. Any concomitant disease or condition that, in the clinical judgment of the treating physician, is likely to prevent the subject from complying with any aspect of the protocol or that may put the subject at unacceptable risk.
- 17. Subjects with  $\geq$  grade 1 peripheral neuropathy at screening.

### 6 Study Drug

### 6.1 Study Drug Administration

<u>Cohorts 1 and 2:</u> For each cycle 1, a single oral dose of IACS-010759 will be administered on day 1. The next dose of IAC-010759 will be administered on day 8, and daily continuously for the duration of the study with no interruptions unless there are adverse events as described in Section 4.1.9. IACS-010759 doses will be separated by intervals of approximately 24 hours (+/- 3 hours).

<u>Cohorts 3-6 and Dose Expansion</u>: Based on the observed accumulation of IACS-010759 throughout the dosing period in cohorts 1 and 2, a modified dosing regimen is being implemented, consisting of an induction phase in which IACS-010759 is administered daily for up to 7 days, followed by a maintenance phase in which a lower dose is administered weekly (or as otherwise specified by the SMC based on safety, PK and PD data observed) to maintain steady state plasma levels. Dosing will proceed on this schedule for the duration of the study with no interruptions unless there are adverse events as described in Section 4.1.9.

IACS-010759 will be administered without food, at least 1 hour before and at least 2 hours after eating. Each dose of IACS-010759 should be administered with 8 ounces of water. If a dose is missed, the next dose will not be increased to account for missing a dose. The subject will take the next regular dose at the scheduled time. Following cycle 1 (28-day cycle for cohorts 1 and 2, 21 day cycle for subsequent cohorts), subjects will receive one cycle of therapy every 21 days (+/- 4 days).

In cohorts 1 and 2, treatment was administered as an inpatient for 24 hours on day 1 and then starting on day 8 for the next 7 days for all enrolled subjects. In cohorts 3 and 4, treatment will be administered as an inpatient for 24 hours on Day 7 of Cycle 1 for all enrolled subjects. In subsequent cohorts, treatment will be administered as an inpatient for 24 hours on Day 5 of Cycle 1 for all enrolled subjects. IACS-010759 will be self-administered and subjects instructed not to dose on days when PK/PD samples are collected until advised by the research staff. Self-administration can occur on days without PK/PD and subjects will record administration in a provided diary.

In the expansion phase, after the first 6 subjects have been enrolled in the expansion cohort, the next 6 subjects will be enrolled in the Food Effect group where the effect of a high fat meal on the PK of IACS-010759 will be evaluated on day 1 of cycle 1 for the cohort (Food Effect group). The dose level to be administered will be the single agent RP2D induction dose as determined in the escalation phase or may be lower than the RP2D if clinical safety concerns prevent the use of RP2D for the food effect evaluation. Subjects in the Food Effect group will consume the high-fat meal within 30 minutes *prior to* IACS-010759 administration and blood samples collected at

the timepoints listed in the Study Flowchart for PK analysis. After this day 1 dose, subsequent doses of IACS-010759 will be administered without food as described above for the remainder of the cycle. The plasma levels in these subjects will be compared to those of the other subjects in the expansion cohort to determine whether consumption of a meal affects the plasma levels of IACS-010759.

### **6.2 Study Drug Information**

MDACC, IACS has defined a chemical synthesis process, specific purity profile and release specifications for the manufacture of IACS-010759. WuXi AppTec Co, Ltd. is producing GMP material on a 2.5 kg scale. The final drug product will be a dry filled capsule (DFC) formulation for oral administration.

Study drug will be packaged in 28-count bottles of 4 strengths: 0.1 mg, 0.5 mg, 1.0 mg and 5.0 mg, as described in Table 6. The first dose strength to be administered in cohort 1 of the dose escalation phase is 0.5 mg. Study drug may be stored at room temperature.

Table 6: IACS-010759 Drug Product Appearance by Strength

| Strength | Appearance |
|---|---|
| 0.1 mg | Hard Gelatin capsules, Size 3, white opaque cap, white opaque body |
| 0.5 mg | Hard Gelatin capsules, Size 3, light green opaque cap, white opaque body |
| 1.0 mg | Hard Gelatin capsules, Size 3, light blue opaque cap, white opaque body |
| 5.0 mg | Hard Gelatin capsules, Size 3, dark blue opaque cap, white opaque body |

The active ingredient in IACS-010579 is manufactured under GMP conditions by: Shanghai SynTheAll Pharmaceutical Co. Ltd., 9 Yuegong Road, Jinshan District, Shanghai 201507, China

The finished drug product is manufactured under GMP conditions by: WuXi AppTec Co., Ltd, 299 FuTe Zhong Road, Waigaoqao Free Trade Zone, Shanghai, 200131, P. R. China

### 6.3 Drug Overdose Management

There are no known antidotes available for the IACS-010759. Any overdoses with this drug should be managed symptomatically.

## 7 Concurrent and Supportive Therapies

### 7.1 Non-Permitted Concomitant Therapies

Subject <u>may not</u> receive the following concomitant therapies during the study:

| 1. | Biguanides or other agents known to increase risk of lactic acidosis (Appendix 10.1) |
|---|---|
| 2. | High dose steroids (>20 mg prednisolone or equivalent per day) including for GVHD |
| 3. | Immunosuppressive drugs with the exception of cyclosporine and tacrolimus |
| 4. | Erythropoietin and growth factors are not permitted to be used prophylactically in cycle 1 but allowed if needed in cycle 2 and onwards. However, these can be used therapeutically throughout the study. |
| 5. | Other cancer therapy (chemotherapy, radiation or immunotherapy) other than the exceptions mentioned in Inclusion Criteria #9. |
| 6. | Strong cytochrome P450 (CYP450) inhibitors or inducers, as specified below: |

| CYP Enzyme | Strong Inhibitors | Strong Inducers |
|---|---|---|
| CYP1A2 | Ciprofloxacin, clinafloxacin, enoxacin, fluvoxamine, zafirlukast | |
| CYP2C8 | Gemfibrozil | |
| CYP2C19 | Fluconazole, fluvoxamine, ticlopidine | |
| СҮРЗА | Clarithromycin, conivaptan, grapefruit juice, itraconazole, ketoconazole, mibefradil, nefazodone, posaconazole, telithromycin, troleandomycin, voriconazole | Avasimibe, carbamazepine, phenobarbital, phenytoin, pioglitazone, rifbatun, rifampin, St. John's wort |
| CYP2D6 | Bupropion, fluoxetine, paroxetine, quinidine | |

### 7.2 Supportive Care Guidelines & Permitted Concomitant Therapies

### 7.2.1 Concomitant medication/therapies

In general, the use of any concomitant medication/therapies deemed necessary for subject supportive care and safety are permitted. Subjects with high WBC counts may receive hydroxyurea prior to study entry and during the first 2 cycles. Concurrent therapy for CNS prophylaxis or continuation of therapy for controlled CNS disease is permitted as defined in the inclusion criteria. With the exception of these agents, concomitant systemic chemotherapy is not permitted.

Concomitant medications are recommended as prophylaxis for nausea, vomiting, and infections, and are allowed for managing myelosuppression as shown in the table below. Concomitant medications will be recorded in the Case Report Form.

IACS2015-001: Protocol Amendment #11 (01-21-20) 

Table 8: Instructions for the use of concomitant medications and therapies

| Category of Use | Medication | Comment on Use | Restriction on Use |
|---|---|---|---|
| Recommended | Prophylactic antibiotics, antifungal agents, and antiviral agents. | Strongly encouraged | Agents known to increase risk of lactic acidosis (see Appendix 10.1) |
| | Antiemetic agents | According to standard of care at MDACC | None |
| Allowed | Oral allopurinol or rasburicase | At investigators discretion | None |
| | Leukapheresis | According to standard of care at MDACC | Before induction 1 day 1 only |
| | Red blood cell transfusion | None | None |
| | Platelet transfusion | None | None |
| | White blood cell transfusion | At investigators discretion according to standard of care at MDACC | None |
| | Myeloid growth factors or platelet growth factor | At investigators discretion according to standard of care at MDACC | None |
| | Erythropoietin or darbepoetin | At investigators discretion according to the standard of care at MDACC | None |
| | Any other medication for supportive care | At investigators<br>discretion according to<br>standard of care at<br>MDACC | Agents known to increase risk of lactic acidosis (see Appendix 10.1) |

### 7.2.2 Use of Blood Products

During the administration of IACS, subjects may receive red blood cell (RBC) or platelet transfusions, if clinically indicated, per institutional guidelines.

Myelosuppression is expected in subjects with AML due to underlying disease. Most subjects will have neutropenia, thrombocytopenia, or both at study entry. Significant or life-threatening myelosuppression may be managed with growth factor support including G-CSF, GM-CSF and platelet growth factors and erythropoietin/darbopoietin/blood transfusion according to institutional standard of care, American Society of Clinical Oncology (ASCO) Practice Guidelines, and/or NCCN Practice Guidelines.

### 7.2.3 Lactic Acidosis and Severe Acidemia Management

Subjects with lactic acidosis and severe acidemia (pH < 7.1) should be seen by a nephrology specialist as soon as possible and receive bicarbonate therapy. When using bicarbonate therapy in subjects with lactic acidosis and severe acidemia, the aim is to maintain the arterial pH above 7.1. Rapid infusions of sodium bicarbonate may increase the pCO<sub>2</sub>, accelerate the production of lactate, lower the ionized calcium, expand the extracellular space, and raise the serum sodium concentration. There is little evidence that any alternative buffering agents are superior to bicarbonate therapy. In adequately ventilated subjects with lactic acidosis and severe acidemia, 1 to 2 mEq/kg sodium bicarbonate is given as an intravenous bolus. This dose is repeated after 30 to 60 minutes if the pH is still below 7.1.

### 8 Administrative, Legal & Ethical Requirements

### 8.1 Adverse Event, serious adverse event and reporting

### 8.1.1 Adverse Event (AE):

Any untoward medical occurrence in a subject or clinical investigation subject administered an investigational product. An AE does not necessarily have a causal relationship with the medicinal product.

The criteria for identifying AEs are:

- Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
- Any new disease or exacerbation of an existing disease
- Any deterioration in non-protocol-required measurements of laboratory value or other clinical test (e.g., ECG or X-ray) that results in symptoms, a change in treatment, or discontinuation from study drug
- Recurrence of an intermittent medical condition (e.g. headache) not present at Baseline.

An abnormal laboratory test result may be considered as an adverse event if the identified laboratory abnormality leads to any type of intervention whether prescribed in the protocol or not.

A laboratory result should be considered by the Investigator to be an adverse event if it:

- Results in the withdrawal of study treatment
- Results in withholding of study treatment pending some investigational outcome
- Medical evaluation, results in the initiation of an intervention (e.g. potassium supplement for hypokalemia)
- Any out of range laboratory value that in the Investigator's judgment, fulfills the definitions of an AE with regards to subject's medical profile
- Increases in severity compared to Baseline by ≥ 2 NCI grades (see Appendix C for NCI CTCAE Ver 4.03 criteria), with the exception of lymphocytes, albumin, cholesterol, glucose and phosphate. For these tests, a change of ≥ 2 grades will be evaluated by the Investigator to determine if they are of clinical significance and if so, will be considered an adverse event.

IACS2015-001: Protocol Amendment #11 (01-21-20) 

Abnormal laboratory values should not be listed as separate AEs if they are considered to be part of the clinical syndrome that is being reported as an AE. Any laboratory abnormality considered to constitute an adverse event should be reported on the Adverse Event Case Report Form (CRF).

It is the responsibility of the Investigator to review all laboratory findings, including laboratory assessments performed at outside labs, in all subjects and determine if they constitute an adverse event. Medical and scientific judgment should be exercised in deciding whether an isolated laboratory abnormality should be classified as an adverse event. The Investigator will assess external laboratory findings and determine clinical significance of any which are deemed adverse events. In these instances, the laboratory reports should be signed and dated by the Investigator.

### **8.1.2** Reporting of Adverse Events

Adverse events will be recorded by the research personnel on the CRF. The Investigator or physician designee is responsible for verifying and providing source documentation for all adverse events and assigning the attribution for each event for all subjects enrolled on the trial.

For this protocol, adverse events and protocol specific data will be entered into the electronic case report form. Serious adverse events will be entered into ARISg and reconciled against the clinical data base at the end of the study. All AEs encountered during the clinical study will be reported on the CRF. All AEs, regardless of relationship to study drug or procedure, should be collected, beginning from the time of the first protocol-specific intervention (study drug administration). New information regarding signs and symptoms that occurred prior to the first study medication dose on Day 1 should be recorded under the subject's Medical History. Adverse events in clinical investigation subjects include any change in the subject's condition. This includes symptoms, physical findings, or clinical syndromes.

Subjects with AEs that are ongoing at the subject's last study visit must be followed until resolution or for 30 days after the subject's last study visit, whichever comes first. Adverse events that are reported during the Follow-up Period will be recorded on the Adverse Events CRF and followed until resolution or for up to the 30 days after the subject's last study visit, whichever comes first, with the exception that SAEs will be followed until the event resolves or the event or sequelae stabilize.

Every effort must be made by the Investigator to categorize each AE according to its severity and its relationship to the study treatment.

#### **8.1.3** Assessing Severity of Adverse Events

The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE Ver 4.03; <a href="http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE">http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE</a> 4.03 2010-06-14 QuickReference 8.5x11.pdf) is used to assign severity scales to AEs.

They are:

Grade 1 = Mild

Grade 2 = Moderate

Grade 3 = Severe

Grade 4 = Life Threatening

Grade 5 = Death

Elevated lactate levels are an anticipated pharmacodynamic effect of OXPHOS inhibitors. It is currently unknown if such effects may lead to biological consequences, such as lactic acidosis or

associated symptoms. Safety and tolerability of IACS-010759 is the primary objective of this phase 1 clinical trial. During this study, if elevated lactate levels are observed and subjects are hospitalized for observation of signs and symptoms (as described in Section 4.1.11), such hospitalization (or prolongation of hospitalization) for observation of signs and symptoms that would not otherwise require hospitalization will not be considered as a grade 3 toxicity when grading the severity of the adverse event if subjects remain asymptomatic and pH remains normal.

In addition, all AEs reported using the NCI CTCAE Ver 4.03 classification and graded as 4 or 5 are to be considered serious. The recommended Adverse Event Recording Guidelines are provided in Section 8.1.7.

The criteria for assessing severity are different than those used for seriousness.

#### 8.1.4 Assessing Relationship to Study Treatment

Items to be considered when assessing the relationship of an AE to the study treatment are:

- Temporal relationship of the onset of the event to the initiation of the study treatment
- The course of the event, considering especially the effect of discontinuation of study treatment or reintroduction of study treatment, as applicable
- Whether the event is known to be associated with the study treatment, or with other similar treatments
- The presence of risk factors in the study subject known to increase the occurrence of the event
- The presence of non-study treatment related factors which are known to be associated with the occurrence of the event

#### 8.1.5 Classification of Causality

**Causality** is a determination of whether there is a reasonable possibility that the drug may have caused or contributed to an adverse event. It includes assessing temporal relationships, dechallenge/rechallenge information, association (or lack of association) with underlying diseases, and the presence (or absence) of one or more likely causes.

The investigator must attempt to determine whether an adverse event is in some way related to the use of the study drug. This relationship should be described as follows:

**Unlikely:** The event is clearly due to causes distinct from the use of the study drug, such as a documented pre-existing condition, the effect of a concomitant medication, or a new condition that, based on the pathophysiology of the condition and the pharmacology of the study drug, is unlikely to be related to the use of the study drug.

**Possible:** The event follows a reasonable temporal sequence from administration of the study drug or the event follows a known response pattern to the study drug, *but* the event could have been produced by a concomitant medication or an intercurrent medical condition which, based on the pathophysiology of the condition and the pharmacology of the study drug, is unlikely to be related to the use of the study drug.

**Probable:** The event follows a reasonable temporal sequence from administration of the study drug and the event follows a known response pattern to the study drug and the event cannot be

reasonably explained by an intercurrent medical condition *or* the event cannot be the effect of a concomitant medication.

**Definite:** The event follows a reasonable temporal sequence from administration of the study drug, the event follows a known response pattern to the study drug, and based on the known pharmacology of the study drug, the event is clearly related to the effect of the study drug.

**Unknown:** Based on the evidence available, causality cannot be ascribed.

### 8.1.6 Reporting Requirements

Reporting requirements will be as per institutional guidelines.

### Adverse events (AE) related to study conditions

The serious adverse event (SAE) reporting period will begin with the time of the first protocol-specific intervention (study drug administration) Regardless of severity or seriousness, new information regarding signs and symptoms that occurred prior to the first study medication dose on Day 1 should be recorded under the subject's Medical History.

AEs should be followed to resolution or stabilization, and reported as SAEs if they become serious. This also applies to subjects experiencing AEs that cause interruption or discontinuation of investigational product, or those experiencing AEs that are present at the end of their participation in the study. Such subjects should receive post-treatment follow-up as appropriate.

### 8.1.7 Serious Adverse Event Reporting (SAE)

An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or the sponsor, it results in any of the following outcomes:

- Death
- A life-threatening adverse drug experience any adverse experience that places the subject, in the view of the initial reporter, at immediate risk of death from the adverse experience as it occurred. It does not include an adverse experience that, had it occurred in a more severe form, might have caused death.
- Subject hospitalization or prolongation of existing hospitalization
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- A congenital anomaly/birth defect.

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon appropriate medical judgment, they may jeopardize the subject or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in subject hospitalization, or the development of drug dependency or drug abuse (21 CFR 312.32).

Important medical events as defined above, may also be considered serious adverse
events. Any important medical event can and should be reported as an SAE if deemed
appropriate by the Principal Investigator or the IND Sponsor, to the PROMETRIKA Safety
Manager.

- All events occurring during the conduct of a protocol and meeting the definition of a SAE must be reported to the IRB in accordance with the timeframes and procedures outlined in "The University of Texas M. D. Anderson Cancer Center Institutional Review Board Policy for Investigators on Reporting Unanticipated Adverse Events for Drugs and Devices". Unless stated otherwise in the protocol, all SAEs, expected or unexpected, must be reported to the PROMETRIKA Safety Manager, regardless of attribution (within 5 working days of knowledge of the event).
- All life-threatening or fatal events, that are unexpected, and related to the study drug, must have a written report submitted within 24 hours (next working day) of knowledge of the event to the PROMETRIKA Safety Project Manager.
- Unless otherwise noted, the entry of an AE that is designated as serious in the EDC system will automatically prompt an automated email alert for a newly entered case or for an existing case where a change in status of the AE fields has been made by the site. The email alert will be sent to relevant personnel involved with the SAE case management, including the PROMETRIKA Safety Manager. In the event that the site is unable to send the information through the EDC, the site will contact the Drug Safety Management department at PROMETRIKA by phone (617.844.0205) or fax (617.868.2122) and forward the SAE Form and other related documents to the PROMETRIKA Safety Manager. The site will be responsible for safety reporting to the MDACC IRB.
- Serious adverse events will be captured from the time of the first protocol-specific
  intervention (study drug administration), until 30 days after the last dose of drug, unless
  the participant withdraws consent. Serious adverse events must be followed until
  clinical recovery is complete and laboratory tests have returned to baseline, progression
  of the event has stabilized, or there has been acceptable resolution of the event.
- Additionally, all serious adverse events that occur after the 30 day time period that are related to the study treatment must be reported to the Sponsor and the PROMETRIKA Safety Manager. This may include the development of a secondary malignancy.

IACS2015-001: Protocol Amendment #11 (01-21-20)

### **Recommended Adverse Event Recording Guidelines**

| | Recommend | ded Adverse | Event Record | ing Guideline | es |
|---|---|---|---|---|---|
| Attribution | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
| , action | | | | | |
| Unrelated | Phase I | Phase I | Phase I<br>Phase II | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III |
| Unlikely | Phase I | Phase I | Phase I<br>Phase II | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III |
| Possible | Phase I<br>Phase II | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III |
| Probable | Phase I<br>Phase II | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III |
| Definitive | Phase I<br>Phase II | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III | Phase I<br>Phase II<br>Phase III |

#### 8.1.8 Reporting to FDA:

PROMETRIKA will submit **all** SAE reports to the IND Office via e-mail to <u>MDACCSafetyReports@mdanderson.org</u>. Serious adverse events will be submitted to FDA by the IND Sponsor (Safety Project Manager, IND Office) according to 21 CFR 312.32.

It is the responsibility of the PI and the research team to ensure serious adverse events are reported according to the Code of Federal Regulations, Good Clinical Practices, the protocol guidelines, the sponsor's guidelines, and Institutional Review Board policy.

### 8.1.9 Unexpected Adverse Event

An unexpected adverse event is one that is not listed in the current Clinical Investigator's Brochure (CIB) / Package Insert or that differs from the event mentioned in the CIB / Package Insert because of greater severity or specificity.

# 9 Appendices

# 9.1 Causes of elevated lactate

| Shock | Pharmacological agents* |
|---|---|
| Distributive | Linezolid |
| Cardiogenic | Nucleoside reverse transcriptase inhibitors |
| Hypovolemic | Metformin |
| Obstructive | Epinephrine |
| Post-cardiac arrest | Propofol |
| Regional tissue ischemia | Acetaminophen |
| Mesenteric ischemia | Beta <sub>2</sub> agonists |
| Limb ischemia | Theophylline |
| Burns | |
| Trauma | Anaerobic muscle activity |
| Compartment syndrome | Seizures |
| Necrotizing soft tissue infections | Heavy exercise |
| Diabetic ketoacidosis | Excessive work of breathing |
| Drugs/toxins | Thiamine deficiency |
| Alcohols | Malignancy |
| Cocaine | Liver failure |
| Carbon monoxide | Mitochondrial disease |
| Cyanide | |

Adapted from [23]

IACS2015-001: Protocol Amendment #11 (01-21-20) 

### 9.2 List of abbreviations

AML Acute Myeloid Leukemia
ANC Absolute Neutrophil Count
CBC Complete Blood Chemistry

CR Complete Remission

CRi Complete Remission with Incomplete Hematological Recovery

CTCAE Common Terminology Criteria for Adverse Events

DDI Drug-drug interaction
DLT Dose-limiting Toxicity

eCRF Electronic Case Report Form

GCP Good Clinical Practice

HI Hematologic Improvement

IACS Institute for Applied Cancer Science

IB Investigator's Brochure
ICF Informed Consent Form

ICH International Conference on Harmonisation

IRB Institutional Review Board

LC-MS Liquid Chromatography—Mass Spectrometry

LSC Leukemic Stem Cells

MDACC MD Anderson Cancer Center MTD Maximum Tolerated Dose

MLFS Morphologic leukemia-free state
NOAEL No Observed Adverse Effect Level

ORR Overall Response Rate
OXPHOS Oxidative Phosphorylation

PD Pharmacodynamic PK Pharmacokinetic

pAMPK Adenosine Monophosphate Activated Protein Kinase

PI Principal Investigator
PR Partial Remission
RD Recurrence of Disease

RP2D Recommended Phase 2 Dose

QTcF Fridericia Correction Formula

SAE Serious Adverse Event
SCT Stem Cell Transplant
SD Standard Deviation
ULN Upper Limit of Normal

### 9.3 ECOG Performance Status\*

| Grade | ECOG |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair |
| 5 | Dead |

<sup>\*</sup> As published in Am. J. Clin. Oncol.: Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982.

# 9.4 New York Heart Association (NYHA) Functional Classification

| Class | Patient Symptoms |
|---|---|
| I | No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath). |
| II | Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath). |
| III | Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea. |
| IV | Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases. |

### 9.5 References

- 1. Siegel, R., D. Naishadham, and A. Jemal, *Cancer statistics, 2013.* CA Cancer J Clin, 2013. **63**(1): p. 11-30.
- 2. Heerema-McKenney, A. and D.A. Arber, *Acute myeloid leukemia*. Hematol Oncol Clin North Am, 2009. **23**(4): p. 633-54.

IACS2015-001: Protocol Amendment #11 (01-21-20) 

- 3. Kadia, T.M., et al., *Toward Individualized Therapy in Acute Myeloid Leukemia: A Contemporary Review.* JAMA Oncol, 2015. **1**(6): p. 820-8.
- 4. Estey, E., Acute myeloid leukemia and myelodysplastic syndromes in older subjects. J Clin Oncol, 2007. **25**(14): p. 1908-15.
- 5. Ravandi, F., et al., *Characteristics and outcome of subjects with acute myeloid leukemia refractory to 1 cycle of high-dose cytarabine-based induction chemotherapy.* Blood, 2010. **116**(26): p. 5818-23; quiz 6153.
- 6. Giles, F., et al., *Outcome of subjects with acute myelogenous leukemia after second salvage therapy.* Cancer, 2005. **104**(3): p. 547-54.
- 7. O'Brien, S., et al., *Outcome of adults with acute lymphocytic leukemia after second salvage therapy.* Cancer, 2008. **113**(11): p. 3186-91.
- 8. Caro, P., et al., *Metabolic signatures uncover distinct targets in molecular subsets of diffuse large B cell lymphoma*. Cancer Cell, 2012. **22**(4): p. 547-60.
- 9. Haq, R., et al., Oncogenic BRAF regulates oxidative metabolism via PGC1alpha and MITF. Cancer Cell, 2013. **23**(3): p. 302-15.
- 10. Muller, F.L., et al., *Passenger deletions generate therapeutic vulnerabilities in cancer.* Nature, 2012. **488**(7411): p. 337-42.
- 11. Roesch, A., et al., *Overcoming intrinsic multidrug resistance in melanoma by blocking the mitochondrial respiratory chain of slow-cycling JARID1B(high) cells.* Cancer Cell, 2013. **23**(6): p. 811-25.
- 12. Vazquez, F., et al., *PGC1alpha expression defines a subset of human melanoma tumors with increased mitochondrial capacity and resistance to oxidative stress.* Cancer Cell, 2013. **23**(3): p. 287-301.
- 13. Viale, A., et al., Oncogene ablation-resistant pancreatic cancer cells depend on mitochondrial function. Nature, 2014. **514**(7524): p. 628-32.
- 14. Birsoy, K., et al., An Essential Role of the Mitochondrial Electron Transport Chain in Cell Proliferation Is to Enable Aspartate Synthesis. Cell, 2015. **162**(3): p. 540-51.
- 15. Lagadinou, E.D., et al., *BCL-2 Inhibition Targets Oxidative Phosphorylation and Selectively Eradicates Quiescent Human Leukemia Stem Cells.* Cell stem cell, 2013.
- 16. Samudio, I., et al., *Pharmacologic inhibition of fatty acid oxidation sensitizes human leukemia cells to apoptosis induction.* The Journal of clinical investigation, 2010. **120**(1): p. 142-56.
- 17. Sriskanthadevan, S., et al., AML cells have low spare reserve capacity in their respiratory chain that renders them susceptible to oxidative metabolic stress. Blood, 2015. **125**(13): p. 2120-30.
- 18. Sullivan, L.B., et al., Supporting Aspartate Biosynthesis Is an Essential Function of Respiration in Proliferating Cells. Cell, 2015. **162**(3): p. 552-63.
- 19. Simsek, T., et al., *The distinct metabolic profile of hematopoietic stem cells reflects their location in a hypoxic niche.* Cell stem cell, 2010. **7**(3): p. 380-90.
- 20. Thall, P.F., R.M. Simon, and E.H. Estey, *Bayesian sequential monitoring designs for single-arm clinical trials with multiple outcomes*. Stat Med, 1995. **14**(4): p. 357-79.
- 21. Kruse, O., N. Grunnet, and C. Barfod, *Blood lactate as a predictor for in-hospital mortality in subjects admitted acutely to hospital: a systematic review.* Scand J Trauma Resusc Emerg Med, 2011. **19**: p. 74.
- 22. Cheson, B.D., et al., Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol, 2003. 21(24): p. 4642-9.

| 23. | Andersen, L.W., et al., <i>Etiology and therapeutic approach to elevated lactate levels</i> . Mayo Clin Proc, 2013. <b>88</b> (10): p. 1127-40. |
|---|---|